CLINICAL TRIAL: NCT00118365
Title: A Phase III Randomized, Double-Blind, Placebo-Controlled Clinical Trial of the Combination of DFMO and Sulindac to Decrease the Rate of Recurrence of Adenomatous Polyps in the Colon
Brief Title: Eflornithine and Sulindac in Preventing Colorectal Cancer in Patients With Colon Polyps
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2009-00880; UCI 97-05; R01CA088078 (NIH); NCT00005882 (obsolete NCT alias)
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Results first posted 2015-01-22 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2014-02

CONDITIONS: Precancerous Condition
MeSH Terms: conditions — Precancerous Conditions | interventions — Eflornithine; Sulindac

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm II (placebo) (Placebo Comparator): Patients receive oral double placebo once daily. In both arms, treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  Interventions: Other: placebo; Other: laboratory biomarker analysis
- Arm I (eflornithine and sulindac) (Experimental): Patients receive oral eflornithine (DFMO) and oral sulindac once daily. In both arms, treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  Interventions: Drug: eflornithine; Drug: sulindac; Other: laboratory biomarker analysis

INTERVENTIONS:
Other: placebo — Given orally
  Other Names: PLCB
  Arms: Arm II (placebo)
Drug: eflornithine — Given orally
  Other Names: 2-difluoromethylornithine; DFMO; difluromethylornithine
  Arms: Arm I (eflornithine and sulindac)
Drug: sulindac — Given orally
  Other Names: Aflodac; Algocetil; Clinoril; SULIN
  Arms: Arm I (eflornithine and sulindac)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase III trial is studying eflornithine and sulindac to see how well they work compared to a placebo in preventing colorectal cancer in patients with colon polyps. Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of eflornithine and sulindac may prevent colorectal cancer. It is not yet known whether eflornithine and sulindac are more effective than a placebo in preventing colorectal cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the rate of new adenomatous polyp formation in patients with a history of adenomatous polyps of the colon treated with eflornithine and sulindac vs placebo.

II. Correlate the effects of eflornithine and sulindac on polyamine and prostaglandin content in the flat mucosa with the rate of new adenoma formation in these patients.

III. Compare the rate of side effects in patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to participating center and aspirin use (yes vs no).

Patients receive oral double placebo once daily for 4 weeks. Patients who are more than 70% compliant by pill measurement or self reporting are randomized to 1 of 2 treatment arms.

Arm I: Patients receive oral double placebo once daily.

Arm II: Patients receive oral eflornithine (DFMO) and oral sulindac once daily.

In both arms, treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.

ELIGIBILITY:
Criteria:

* History of >= 1 surgically resected adenomatous polyp of the colon measuring >= 3 mm within the past 5 years
* Screening colonoscopy performed within the past 6 months
* All polyps must have been removed during colonoscopy, pathologically examined, and archived
* No prior surgical resection removing > 40 cm of the colon
* No personal or family history of familial polyposis or hereditary non-polyposis colon cancer
* SWOG 0-1
* Bilirubin =< 2.0 mg/dL
* AST and ALT =< 2 times normal
* Creatinine =< 1.5 mg/dL
* Urine protein =<, urine casts 0-3, urine WBC and RBC count 0-5 cells by urinalysis
* No history of inflammatory bowel disease
* No gastric or duodenal ulcers within the past 12 months
* Gastric or duodenal ulcers that were adequately treated > 24 months ago are allowed
* No symptomatic gastric or duodenal ulcers
* Not pregnant or nursing
* Negative pregnancy test
* Must have regional geographic stability over the next 36 months
* Pure tone audiometry evaluation normal
* Patients with >= 20 dB of uncorrectable hearing loss (for age) of any 2 contiguous frequencies are not allowed
* No invasive malignancy within the past 5 years except adequately treated nonmelanoma skin cancer, level I (or Breslow < 0.76 mm) cutaneous melanoma, Duke's A colon cancer, stage I cervical cancer, or stage 0 chronic lymphocytic leukemia
* No severe metabolic disorder
* No other significant acute or chronic disease that would preclude study participation
* No history of abnormal wound healing or repair
* No conditions that would confer risk of abnormal wound healing or repair
* No history of allergy to NSAIDs or eflornithine
* No concurrent chemotherapy
* No concurrent corticosteroids on a regular or predictable intermittent basis
* No concurrent radiotherapy
* Concurrent calcium supplements (=< 1,000 mg/day) allowed
* Concurrent lipid-lowering drugs (i.e., high-dose statins) allowed
* No other concurrent nonsteroidal anti-inflammatory drugs (NSAIDs) on a regular or predictable intermittent basis
* Concurrent aspirin for cardiovascular prophylaxis (i.e., 81 mg/day) allowed
* No concurrent anticoagulants on a regular or predictable intermittent basis
* No concurrent treatment for gastric or duodenal ulcers

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 1998-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Meyskens, Principal Investigator — University of California Medical Center At Irvine-Orange Campus
Locations (1):
- University of California Medical Center At Irvine-Orange Campus, Orange, California, United States

REFERENCES:
- [Derived] Thompson PA, Wertheim BC, Zell JA, Chen WP, McLaren CE, LaFleur BJ, Meyskens FL, Gerner EW. Levels of rectal mucosal polyamines and prostaglandin E2 predict ability of DFMO and sulindac to prevent colorectal adenoma. Gastroenterology. 2010 Sep;139(3):797-805, 805.e1. doi: 10.1053/j.gastro.2010.06.005. Epub 2010 Jun 9. PMID 20538001

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Eflornithine and Sulindac) | Arm II (Placebo)
Started | 191 | 184
Completed | 132 | 124
Not Completed | 59 | 60

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Eflornithine and Sulindac) | Arm II (Placebo) | Total
Number analyzed (Participants) | 191 | 184 | 375
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (8.6) | 61 (8.4) | 60.5 (8.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 46 | 90
  Male | 147 | 138 | 285

OUTCOME MEASURES:

1. Primary Outcome: Detection of Any Adenoma at the End of the Study
Description: Detection of any adenoma at the end of the study. This analysis is based on the participants who had the end-of-study colonscopy procedure done.
Time Frame: Up to 36 months
Population: This analysis is based on the participants who had the end-of-study colonscopy procedure done.
Measure: Number; unit: participants
Arm/Group | Arm I (Eflornithine and Sulindac) | Arm II (Placebo)
Number analyzed (Participants) | 138 | 129
participants
  Yes | 17 | 53
  No | 121 | 76

2. Secondary Outcome: Detection of Any Adenoma at the End of the Study Stratified by Baseline Prostaglandin E2 (PGE2) and Treatment
Description: This analysis is based on the participants who had the end-of-study colonscopy procedure done and their baseline PGE2 values are available. The low PGE2 is defined as the values that are below the median PGE2 value in the analysis cohort. The high PGE2 is defined as the values that are above the median PGE2 value in the analysis cohort.
Time Frame: Up to 36 months
Population: This analysis is based on the participants who had the end-of-study colonscopy procedure done and their baseline PGE2 values are available. The low PGE2 is defined as the values that are below the median PGE2 value in the analysis cohort. The high PGE2 is defined as the values that are above the median PGE2 value in the analysis cohort.
Measure: Number; unit: participants
Groups:
- Eflornithine and Sulindac + Low PGE2 at Baseline: Patients receive oral eflornithine (DFMO) and oral sulindac once daily. The treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  eflornithine: Given orally
  sulindac: Given orally
  laboratory biomarker analysis: Correlative studies
  baseline PGE2 values is below the median
- Eflornithine and Sulindac + High PGE2 at Baseline: Patients receive oral eflornithine (DFMO) and oral sulindac once daily. The treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  eflornithine: Given orally
  sulindac: Given orally
  laboratory biomarker analysis: Correlative studies
  baseline PGE2 values is above the median
- Placebo + Low PGE2 at Baseline: Patients receive oral double placebo once daily. In both arms, treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  placebo: Given orally
  laboratory biomarker analysis: Correlative studies
  baseline PGE2 value is below median
- Placebo + High PGE2 at Baseline: Patients receive oral double placebo once daily. In both arms, treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  placebo: Given orally
  laboratory biomarker analysis: Correlative studies
  baseline PGE2 value is above median
Arm/Group | Eflornithine and Sulindac + Low PGE2 at Baseline | Eflornithine and Sulindac + High PGE2 at Baseline | Placebo + Low PGE2 at Baseline | Placebo + High PGE2 at Baseline
Number analyzed (Participants) | 53 | 44 | 42 | 53
participants
  Yes | 12 | 3 | 19 | 21
  No | 41 | 41 | 23 | 32

3. Secondary Outcome: Detection of Any Adenoma at the End of the Study Stratified by Baseline Putrescine and Treatment
Description: The low is defined as the values that are below the median putrescine level in the analysis cohort. The high is defined as the values that are above the median putrescine level in the analysis cohort.
Time Frame: Up 36 months
Population: In the finalized datasaet, the total number of adnoma detected in the placebo group is 55. The descrepancy in the total number of adnoma detected in placebo group between Outcome Measure 1 and this oucome is due to the revolution of the datatset. The analysis cohort is based on the participants whose data are available and complete.
Measure: Number; unit: participants
Groups:
- Eflornithine and Sulindac + Low Putrescine at Baseline: Patients receive oral eflornithine (DFMO) and oral sulindac once daily. The treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  eflornithine: Given orally
  sulindac: Given orally
  laboratory biomarker analysis: Correlative studies
  baseline Putrescine values is below the median
- Eflornithine and Sulindac + High Putrescine at Baseline: Patients receive oral eflornithine (DFMO) and oral sulindac once daily. The treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  eflornithine: Given orally
  sulindac: Given orally
  laboratory biomarker analysis: Correlative studies
  baseline Putrescine values is above the median
- Placebo + Low Putrescine at Baseline: Patients receive oral double placebo once daily. In both arms, treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  placebo: Given orally
  laboratory biomarker analysis: Correlative studies
  baseline Putrescine value is below median
- Placebo + High Putrescine at Baseline: Patients receive oral double placebo once daily. In both arms, treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  placebo: Given orally
  laboratory biomarker analysis: Correlative studies
  baseline Putrescine value is above median
Arm/Group | Eflornithine and Sulindac + Low Putrescine at Baseline | Eflornithine and Sulindac + High Putrescine at Baseline | Placebo + Low Putrescine at Baseline | Placebo + High Putrescine at Baseline
Number analyzed (Participants) | 70 | 66 | 62 | 67
participants
  Yes | 7 | 10 | 24 | 31
  No | 63 | 56 | 38 | 36

4. Secondary Outcome: Detection of Any Adenoma at the End of the Study Stratified by Baseline Spermidine-to-spermine Ratio and Treatment
Description: The low is defined as the ratios that are below the median spermidine-to-spermine ratio in the analysis cohort. The high is defined as the ratios that are above the median spermidine-to-spermine ratio in the analysis cohort.
  In the finalized datasaet, the total number of adnoma detected in the placebo group is 55. The descrepancy in the total number of adnoma detected in placebo group between Outcome Measure 1 and this oucome is due to the revolution of the datatset.
  The analysis cohort is based on the participants whose data are available and complete.
Time Frame: Up 36 months
Population: as for outcome 3
Measure: Number; unit: participants
Groups:
- Eflornithine and Sulindac + Low Spd:Spm at Baseline: Patients receive oral eflornithine (DFMO) and oral sulindac once daily. The treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  eflornithine: Given orally
  sulindac: Given orally
  laboratory biomarker analysis: Correlative studies
  baseline spermidine-to-spermine ratio is below the median
- Eflornithine and Sulindac + High Spd:Spm at Baseline: Patients receive oral eflornithine (DFMO) and oral sulindac once daily. The treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  eflornithine: Given orally
  sulindac: Given orally
  laboratory biomarker analysis: Correlative studies
  baseline spermidine-to-spermine ratio is above the median
- Placebo + Low Spd:Spm at Baseline: Patients receive oral double placebo once daily. In both arms, treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  placebo: Given orally
  laboratory biomarker analysis: Correlative studies
  baseline spermidine-to-spermine ratio is below median
- Placebo + High Spd:Spm at Baseline: Patients receive oral double placebo once daily. In both arms, treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  placebo: Given orally
  laboratory biomarker analysis: Correlative studies
  baseline spermidine-to-spermine ratio is above median
Arm/Group | Eflornithine and Sulindac + Low Spd:Spm at Baseline | Eflornithine and Sulindac + High Spd:Spm at Baseline | Placebo + Low Spd:Spm at Baseline | Placebo + High Spd:Spm at Baseline
Number analyzed (Participants) | 64 | 72 | 68 | 61
participants
  Yes | 5 | 12 | 31 | 24
  No | 59 | 60 | 37 | 37

5. Secondary Outcome: Detection of Any Adenoma at the End of the Study Stratified by Prostaglandin E2 (PGE2) Response and Treatment
Description: PGE2 Responder = PGE2 values at 36-month are decreased by >=30% in PGE2 values from baseline PGE2 nonresponder = PGE2 values at 36-month are increased, or decreased by < 30% from baseline The analysis cohort is based on the participants whose data are available and complete.
Time Frame: Up to 36 months
Population: The analysis cohort is based on the participants whose data are available and complete.
Measure: Number; unit: participants
Groups:
- Eflornithine and Sulindac + PGE2 Responders: Patients receive oral eflornithine (DFMO) and oral sulindac once daily. The treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  eflornithine: Given orally
  sulindac: Given orally
  laboratory biomarker analysis: Correlative studies
  PGE2 Responder = PGE2 values at 36-month are decreased by >=30% in PGE2 values from baseline
- Eflornithine and Sulindac + PGE2 Nonresponders: Patients receive oral eflornithine (DFMO) and oral sulindac once daily. The treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  eflornithine: Given orally
  sulindac: Given orally
  laboratory biomarker analysis: Correlative studies
  PGE2 nonresponder = PGE2 values at 36-month are increased, or decreased by < 30% from baseline
- Placebo + PGE2 Responders: Patients receive oral double placebo once daily. In both arms, treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  placebo: Given orally
  laboratory biomarker analysis: Correlative studies
  PGE2 Responder = PGE2 values at 36-month are decreased by >=30% in PGE2 values from baseline
- Placebo + PGE2 Nonresponders: Patients receive oral double placebo once daily. In both arms, treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  placebo: Given orally
  laboratory biomarker analysis: Correlative studies
  PGE2 nonresponder = PGE2 values at 36-month are increased, or decreased by < 30% from baseline
Arm/Group | Eflornithine and Sulindac + PGE2 Responders | Eflornithine and Sulindac + PGE2 Nonresponders | Placebo + PGE2 Responders | Placebo + PGE2 Nonresponders
Number analyzed (Participants) | 11 | 35 | 17 | 32
participants
  Yes | 1 | 8 | 4 | 15
  No | 10 | 27 | 13 | 17

6. Secondary Outcome: Detection of Any Adenoma at the End of the Study Stratified by Putrescine Response and Treatment
Description: Putrescine responder = Putrescine values at 36-month are decreased by >=30% from baseline Putrescine nonresponder = Putrescine values at 36-month are increased, or decreased by < 30% from baseline The analysis cohort is based on the participants whose data are available and complete.
Time Frame: Up to 36 months
Population: The analysis cohort is based on the participants whose data are available and complete.
Measure: Number; unit: participants
Groups:
- Eflornithine and Sulindac + Putrescine Responders: Patients receive oral eflornithine (DFMO) and oral sulindac once daily. The treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  eflornithine: Given orally
  sulindac: Given orally
  laboratory biomarker analysis: Correlative studies
  Putrescine responder = Putrescine values at 36-month are decreased by >=30% from baseline
- Eflornithine and Sulindac + Putrescine Nonresponders: Patients receive oral eflornithine (DFMO) and oral sulindac once daily. The treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  eflornithine: Given orally
  sulindac: Given orally
  laboratory biomarker analysis: Correlative studies
  Putrescine nonresponder = Putrescine values at 36-month are increased, or decreased by < 30% from baseline
- Placebo + Putrescine Responders: Patients receive oral double placebo once daily. In both arms, treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  placebo: Given orally
  laboratory biomarker analysis: Correlative studies
  Putrescine responder = Putrescine values at 36-month are decreased by >=30% from baseline
- Placebo + Putrescine Nonresponders: Patients receive oral double placebo once daily. In both arms, treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  placebo: Given orally
  laboratory biomarker analysis: Correlative studies
  Putrescine nonresponder = Putrescine values at 36-month are increased, or decreased by < 30% from baseline
Arm/Group | Eflornithine and Sulindac + Putrescine Responders | Eflornithine and Sulindac + Putrescine Nonresponders | Placebo + Putrescine Responders | Placebo + Putrescine Nonresponders
Number analyzed (Participants) | 61 | 60 | 46 | 72
participants
  Yes | 9 | 7 | 22 | 28
  No | 52 | 53 | 24 | 44

7. Secondary Outcome: Detection of Any Adenoma at the End of the Study Stratified by Spermidine-to-spermine Ratio Response and Treatment
Description: Spermidine-to-spermine ratio responder = ratios at 36-month are decreased by >=30% from baseline Spermidine-to-spermine ratio nonresponder = ratios at 36-month are increased, or decreased by < 30% from baseline The analysis cohort is based on the participants whose data are available and complete.
Time Frame: Up to 36 months
Population: The analysis cohort is based on the participants whose data are available and complete.
Measure: Number; unit: participants
Groups:
- Eflornithine and Sulindac + Spd:Spm Responders: Patients receive oral eflornithine (DFMO) and oral sulindac once daily. The treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  eflornithine: Given orally
  sulindac: Given orally
  laboratory biomarker analysis: Correlative studies
  Spd:Spm Responder = spermidine-to-spermine ratio at 36-month are decreased by >=30% from baseline
- Eflornithine and Sulindac + Spd:Spm Nonresponders: Patients receive oral eflornithine (DFMO) and oral sulindac once daily. The treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  eflornithine: Given orally
  sulindac: Given orally
  laboratory biomarker analysis: Correlative studies
  Spd:Spm nonresponder = spermidine-to-spermine ratio at 36-month increased, or decreased by < 30% from baseline
- Placebo + Spd:Spm Responders: Patients receive oral double placebo once daily. In both arms, treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  placebo: Given orally
  laboratory biomarker analysis: Correlative studies
  SpSpd:Spm Responder = spermidine-to-spermine ratio at 36-month are decreased by >=30% from baseline
- Placebo + Spd:Spm Nonresponders: Patients receive oral double placebo once daily. In both arms, treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  placebo: Given orally
  laboratory biomarker analysis: Correlative studies
  Spd:Spm nonresponder = spermidine-to-spermine ratio at 36-month increased, or decreased by < 30% from baseline
Arm/Group | Eflornithine and Sulindac + Spd:Spm Responders | Eflornithine and Sulindac + Spd:Spm Nonresponders | Placebo + Spd:Spm Responders | Placebo + Spd:Spm Nonresponders
Number analyzed (Participants) | 83 | 38 | 41 | 77
participants
  Yes | 8 | 8 | 17 | 33
  No | 75 | 30 | 24 | 44

8. Secondary Outcome: Adverse Events With a Grade of 3 and Above
Description: Participants reported at least 1 adverse event with a grade of 3 and above, regardless if the event is defined as serious per protocol or other.
  Per protocol, not all grade 3 events are considered as serious events.
Time Frame: Up to 36 months
Measure: Number; unit: participants
Arm/Group | Arm I (Eflornithine and Sulindac) | Arm II (Placebo)
Number analyzed (Participants) | 191 | 184
participants | 46 | 37

9. Secondary Outcome: Baseline Putrescine by ODC Genotype
Description: ODC genotype is the genotype of single nucleotide polymorphisms (SNP) in the ornithine decarboxylase (ODC) promoter The analysis cohort is based on the participants whose data are available and complete.
Time Frame: Baseline
Population: The analysis cohort is based on the participants whose data are available and complete.
Measure: Median (Full Range); unit: nmol/mg protein
Groups:
- ODC1 AA/GA: Patients with AA or GA genotype
- ODC1 GG: Patients with GG genotype
Arm/Group | ODC1 AA/GA | ODC1 GG
Number analyzed (Participants) | 101 | 125
nmol/mg protein | 0.47 [0.01 to 4.60] | 0.56 [0.01 to 5.29]

10. Secondary Outcome: Baseline Spermidine by ODC Genotype
Description: as for outcome 9
Time Frame: Baseline
Population: The analysis cohort is based on the participants whose data are available and complete.
Measure: Median (Full Range); unit: nmol/mg protein
Arm/Group | ODC1 AA/GA | ODC1 GG
Number analyzed (Participants) | 101 | 125
nmol/mg protein | 1.99 [0.76 to 9.18] | 2.17 [1.05 to 8.97]

11. Secondary Outcome: Baseline Spermine by ODC Genotype
Description: as for outcome 9
Time Frame: Baseline
Population: The analysis cohort is based on the participants whose data are available and complete.
Measure: Median (Full Range); unit: nmol/mg protein
Arm/Group | ODC1 AA/GA | ODC1 GG
Number analyzed (Participants) | 101 | 125
nmol/mg protein | 6.82 [2.29 to 19.86] | 7.29 [2.72 to 22.85]

12. Secondary Outcome: At the End of the Study - Putrescine Response by ODC Genotype
Description: Putrescine responder was defined as (tissue putrescine value at baseline - tissue putrescine value at the end of the study)/(tissue putrescine value at baseline) ≥ the threshold. Putrescine non-responder was defined as (tissue putrescine value at baseline - tissue putrescine value at the end of the study)/(tissue putrescine value at baseline) < the threshold. The thresholds range from 0.25 to 0.45 with an increment of 0.5. The below data are shown for the threshold of 0.30.
  ODC genotype is the genotype of single nucleotide polymorphisms (SNP) in the ornithine decarboxylase (ODC) promoter The analysis cohort is based on the participants whose data are available and complete.
Time Frame: At the end of the study
Population: The analysis cohort is based on the participants whose data are available and complete.
Measure: Number; unit: participants
Groups:
- DFMO + Sulindac - GG: Patients with GG genotype receive oral eflornithine (DFMO) and oral sulindac once daily. In both arms, treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  eflornithine: Given orally
  sulindac: Given orally
  laboratory biomarker analysis: Correlative studies
- DFMO + Sulindac - AA/GA: Patients with AA or GA genotype receive oral eflornithine (DFMO) and oral sulindac once daily. In both arms, treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  eflornithine: Given orally
  sulindac: Given orally
  laboratory biomarker analysis: Correlative studies
- Placebo - GG: Patients with GG genotype receive oral double placebo once daily. In both arms, treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  placebo: Given orally
  laboratory biomarker analysis: Correlative studies
- Placebo - AA/GA: Patients with AA or GA genotype receive oral double placebo once daily. In both arms, treatment continues for 36 months in the absence of unacceptable toxicity or the development of an invasive malignancy.
  placebo: Given orally
  laboratory biomarker analysis: Correlative studies
Arm/Group | DFMO + Sulindac - GG | DFMO + Sulindac - AA/GA | Placebo - GG | Placebo - AA/GA
Number analyzed (Participants) | 58 | 40 | 43 | 49
participants
  Responder | 26 | 21 | 12 | 12
  Non-Responder | 32 | 19 | 31 | 37

13. Secondary Outcome: At the End of the Study - Spermidine Response by ODC Genotype
Description: Spermidine responder was defined as (tissue spermidine value at baseline - tissue spermidine value at the end of the study)/(tissue spermidine value at baseline) ≥ the threshold. Spermidine non-responder was defined as (tissue spermidine value at baseline - tissue spermidine value at the end of the study)/(tissue spermidine value at baseline) < the threshold. The thresholds range from 0.25 to 0.45 with an increment of 0.5. The below data are shown for the threshold of 0.30.
  ODC genotype is the genotype of single nucleotide polymorphisms (SNP) in the ornithine decarboxylase (ODC) promoter The analysis cohort is based on the participants whose data are available and complete.
Time Frame: At the end of the study
Population: The analysis cohort is based on the participants whose data are available and complete.
Measure: Number; unit: participants
Arm/Group | DFMO + Sulindac - GG | DFMO + Sulindac - AA/GA | Placebo - GG | Placebo - AA/GA
Number analyzed (Participants) | 58 | 40 | 43 | 49
participants
  Responder | 25 | 12 | 15 | 11
  Non-Responder | 32 | 28 | 28 | 38

14. Secondary Outcome: At the End of the Study - Spermine Response by ODC Genotype
Description: Spermine responder was defined as (tissue spermine value at baseline - tissue spermine value at the end of the study)/(tissue spermine value at baseline) ≥ the threshold. Spermine non-responder was defined as (tissue spermine value at baseline - tissue spermine value at the end of the study)/(tissue spermine value at baseline) < the threshold. The thresholds range from 0.25 to 0.45 with an increment of 0.5. The below data are shown for the threshold of 0.30.
  ODC genotype is the genotype of single nucleotide polymorphisms (SNP) in the ornithine decarboxylase (ODC) promoter The analysis cohort is based on the participants whose data are available and complete.
Time Frame: At the end of the study
Population: The analysis cohort is based on the participants whose data are available and complete.
Measure: Number; unit: participants
Arm/Group | DFMO + Sulindac - GG | DFMO + Sulindac - AA/GA | Placebo - GG | Placebo - AA/GA
Number analyzed (Participants) | 58 | 40 | 43 | 49
participants
  Responder | 7 | 7 | 18 | 10
  Non-Responder | 51 | 33 | 25 | 39

15. Secondary Outcome: Number of Participants Have Adenoma Recurrence in Each ODC1 Genotytpe by Treatment Group
Description: as for outcome 9
Time Frame: Up to 36 months
Population: The analysis cohort is based on the participants whose data are available and complete.
Measure: Number; unit: participants
Arm/Group | DFMO + Sulindac - GG | DFMO + Sulindac - AA/GA | Placebo - GG | Placebo - AA/GA
Number analyzed (Participants) | 64 | 42 | 44 | 53
participants | 7 | 9 | 22 | 18

16. Secondary Outcome: Biomarker in Adenoma: Apoptosis
Description: Apoptosis expression was assessed using cytoplasmic staining. The definitions for the category level for the Apoptosis are: 1. focal (less than 10% cells that are positively stained); 2. less than 50% cells are positively stained; 3. more than 50% cells are positively stained.
Time Frame: At the end of the study
Population: The analysis cohort is based on the participants whose data are available.
Measure: Number; unit: adenoma
Units Other Than Participants: adenoma
Arm/Group | Arm I (Eflornithine and Sulindac) | Arm II (Placebo)
Number analyzed (Participants) | 11 | 38
Number analyzed (adenoma) | 12 | 60
adenoma
  A pattern equal to normal mucosa | 2 | 4
  1.focal (<10%) | 7 | 20
  2.cyto less than 50% | 1 | 23
  3.cyto more than 50% | 2 | 13

17. Secondary Outcome: Biomarker in Adenoma - Ki-67
Description: Estimated mean percent of cells staining postivie for the Ki-67 based on the GEE approach with adjustment for covariates
Time Frame: At the end of the study
Population: The analysis cohort is based on the participants whose data are available.
Measure: Mean (95% Confidence Interval); unit: percentage of cells that are positive
Arm/Group | Arm I (Eflornithine and Sulindac) | Arm II (Placebo)
Number analyzed (Participants) | 11 | 40
percentage of cells that are positive | 59.5 [48.10 to 71.02] | 63.9 [57.35 to 70.39]

18. Secondary Outcome: Biomarker in Adenoma: CEA
Description: carcino-embryonic antigen (CEA) is adenocarcinoma tissue marker that is expressed during adenoma formation.
Time Frame: At the end of the study
Population: The analysis cohort is based on the participants whose data are available.
Measure: Number; unit: Adenoma
Units Other Than Participants: Adenoma
Arm/Group | Arm I (Eflornithine and Sulindac) | Arm II (Placebo)
Number analyzed (Participants) | 11 | 40
Number analyzed (Adenoma) | 12 | 66
Adenoma
  A pattern equal to normal mucosa | 1 | 5
  1.<50% of cells showed staining | 5 | 15
  2.50-90% of cells showed staining | 6 | 35
  3.>90% of cells showed staining | 0 | 9
  Insufficient tissue | 0 | 2

19. Secondary Outcome: Biomarker in Adenoma: Sialyl-TN (B72.3)
Description: sialyl-Tn (B72.3) is adenocarcinoma tissue marker that is expressed during adenoma formation.
Time Frame: At the end of the study
Population: The analysis cohort is based on the participants whose data are available.
Measure: Number; unit: Adenoma
Units Other Than Participants: Adenoma
Arm/Group | Arm I (Eflornithine and Sulindac) | Arm II (Placebo)
Number analyzed (Participants) | 11 | 40
Number analyzed (Adenoma) | 12 | 66
Adenoma
  a pattern equal to normal mucosa | 3 | 11
  1.<10% of the cells in the adenoma showed staining | 7 | 32
  2.10-50% cells showed staining | 2 | 17
  3.>50% cells showed staining | 0 | 5
  Insufficient tissue | 0 | 1

20. Secondary Outcome: Biomarker in Adenoma - p53
Description: Estimated mean percent of cells staining postivie for p53 based on GEE approach with adjument for covariates.
  Tumor protein p53, also known as p53, cellular tumor antigen p53, phosphoprotein p53, or tumor suppressor p53, is a protein that in humans is encoded by the TP53 gene.
Time Frame: At the end of the study
Population: The analysis cohort is based on the participants whose data are available.
Measure: Mean (95% Confidence Interval); unit: percentage of cells that are positive
Arm/Group | Arm I (Eflornithine and Sulindac) | Arm II (Placebo)
Number analyzed (Participants) | 11 | 40
percentage of cells that are positive | 75.6 [51.10 to 100.09] | 70.3 [61.86 to 78.69]

21. Secondary Outcome: Biomarker in Adenoma: Bcl-2
Description: bcl-2 is the anti-apoptotic protein BCL2
Time Frame: At the end of the study, up to 3 years
Population: The analysis cohort is based on the participants whose data are available.
Measure: Number; unit: Adenoma
Units Other Than Participants: Adenoma
Arm/Group | Arm I (Eflornithine and Sulindac) | Arm II (Placebo)
Number analyzed (Participants) | 11 | 40
Number analyzed (Adenoma) | 12 | 66
Adenoma
  A pattern equal to normal mucosa | 4 | 17
  1.<10% of the cells in the adenoma showed staining | 4 | 25
  2.10-50% cells showed staining | 3 | 14
  3.>50% cells showed staining | 1 | 8
  Insufficient tissue | 0 | 2

ADVERSE EVENTS:
Time Frame: The adverse event onset date occurred between the date of run-in and the date of off-study or date of follow-up (up to 3.5 years), when available.
Arm/Group | Arm I (Eflornithine and Sulindac) | Arm II (Placebo)
Serious Adverse Events (participants affected / at risk) | 41/191 | 28/184
Other Adverse Events (participants affected / at risk) | 173/191 | 154/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Eflornithine and Sulindac) (N=191) | Arm II (Placebo) (N=184)
ABDOMINAL PAIN MOST LIKELY SECONDARY TO ACUTE CHOLECYSTITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2) | 0 (0)
ACUTE SHORTNESS OF BREATH R/T CHF, IMPROVED (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ACUTE SHORTNESS OF BREATH; CAD; UNSTABLE ANGINA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ANEURYSM (Cardiac disorders) | 1 (1) | 0 (0)
ANGINA (Cardiac disorders) | 0 (0) | 1 (1)
AORTIC STENOSIS (Cardiac disorders) | 1 (1) | 0 (0)
ARRYTHMIA SINUS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
BASAL CELL CARCINOMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
BENIGN POSITIONAL VERTIGO (Nervous system disorders) | 0 (0) | 1 (1)
BIPOLAR, EXACERBATED (Psychiatric disorders) | 1 (1) | 0 (0)
BLADDER PROLAPSE (Renal and urinary disorders) | 0 (0) | 1 (1)
BROKEN RIGHT TIBIA UNDER KNEE D/T MVA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CARCINOMA PROSTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CELLULITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
CELLULITIS OF RIGHT LEG (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (1)
CHEST PAIN (Cardiac disorders) | 2 (2) | 1 (1)
CHEST PAIN AND PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0)
CHEST PAIN X 3 WKS, R/O CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
COLITIS PSEUDOMEMBRANOUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONGESTIVE HEART FAILURE (Cardiac disorders) | 2 (2) | 0 (0)
COPD EXACERBATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 3 (3) | 0 (0)
CORONARY ARTERY DISEASE POST NON-ST ELEVATION MI (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY ARTERY DISORDER (Cardiac disorders) | 0 (0) | 1 (2)
DEPRESSION SUICIDAL (Psychiatric disorders) | 0 (0) | 1 (1)
DISCHARGE SUMMARY 1/27/02 NEW ONSET ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
DIVERTICULITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
DUCTAL LEFT BREAST CANCER (Reproductive system and breast disorders) | 0 (0) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
FX (L) ELBOW (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
GALLSTONES, PANCREATITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL BLEEDING (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL BLEEDING SECONDARY TO ACUTE GASTROENTERITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI BLEED R/T DIVERTICULA (Gastrointestinal disorders) | 1 (1) | 0 (0)
HEART DISEASE: A. CORONARY, B. NON-Q-WAVE INFARCTION, C. UNSTABLE ANGINA; CORONARY STENTING (Cardiac disorders) | 1 (1) | 0 (0)
HOSPITALIZATION - OVERNIGHT OBSERVATION; LEFT KIDNEY BIOPSY (Renal and urinary disorders) | 1 (1) | 0 (0)
HOSPITALIZATION FOR PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HOSPITALIZATION UTI (Renal and urinary disorders) | 1 (1) | 0 (0)
HOSPITALIZATION VAGINAL BLEEDING TOTAL HYSTERECTOMY (Reproductive system and breast disorders) | 1 (1) | 0 (0)
HOSPITALIZATION; APPENDICITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
HOSPITALIZATION; BENIGN PROSTATIC HYPERTROPHY; ADMITTED FOR TRANSURETHRAL RESECTION OF THE PROSTATE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
HOSPITALIZATION; FRACTURE OF LEFT ANKLE REQUIRING SURGICAL INTERVENTION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HOSPITALIZED FOR ELECTIVE BLADDER SURGERY TO EVALUATE INCONTINENCE AND BIOPSY POSSIBLE TUMOR. (Renal and urinary disorders) | 0 (0) | 1 (1)
INFARCT MYOCARDIAL (Cardiac disorders) | 1 (1) | 0 (0)
INTESTINAL ILEUS STATUS POST CHOLECYSTECTOMY (Gastrointestinal disorders) | 0 (0) | 1 (1)
JOINT DISORDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
KIDNEY CALCULUS (Renal and urinary disorders) | 1 (1) | 0 (0)
LEFT LEG CELLULITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
LEFT URETERAL STONES, OBSTRUCTING (Reproductive system and breast disorders) | 1 (1) | 0 (0)
LUMBAR HERNIATED DISC AND LUMBAR RADICULOPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MALIGNANT EPITHELOID NEOPLASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
MENTAL AND PHYSICAL BREAKDOWN (Psychiatric disorders) | 1 (1) | 0 (0)
MVA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION/CHEST PAIN, ABNORMAL CARDIAC ENZYMES (Cardiac disorders) | 1 (1) | 0 (0)
NEPHROPATHY TOXIC (Renal and urinary disorders) | 0 (0) | 1 (1)
OBSTRUCCTIVE JAUNDICE (Gastrointestinal disorders) | 1 (1) | 0 (0)
PAIN CHEST (Cardiac disorders) | 0 (0) | 1 (1)
PANCREATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PANCREATITIS (Infections and infestations) | 1 (2) | 1 (1)
PARATHYROID DISORDER (Endocrine disorders) | 1 (1) | 0 (0)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMONIA, SEPSIS SYNDROME, ACUTE RENAL FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMONIA; POSSIBLE COPD EXACERBATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PROBABLE RIGHT SUBCORTICAL INFARCT (Nervous system disorders) | 1 (1) | 0 (0)
PROLAPSED CYSTOCELE; TOTAL HYSTERECTOMY WITH BILATERAL SALPINGO-OOPHORECTOMY (Reproductive system and breast disorders) | 1 (1) | 0 (0)
PROSTATE CANCER (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PT WAS IN A MOTOR VEHICLE ACCIDENT…RECEIVED CONTUSIONS AND EXPERIENCED HEAD PAIN. PT WAS RESTRAINED. (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PT. ADMITTED TO HOSPITAL FOR SPIGELIAN HERNIA REPAIR (Gastrointestinal disorders) | 0 (0) | 1 (1)
QUADRUPLE BYPASS SURGERY FOR CAD, UNSTABLE ANGINA (Cardiac disorders) | 1 (1) | 0 (0)
R/O MI (Cardiac disorders) | 0 (0) | 1 (1)
RENAL CYST (Gastrointestinal disorders) | 0 (0) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 1 (1)
RIGHT HIP PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
RIGHT KNEE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
S/P LEFT TOTAL HIP ARTHROSCOPY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SEIZURE ACTIVITY SECONDARY TO CEREBRAL ATROPHY OF RIGHT TEMPORAL LOBE (Nervous system disorders) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
STERNAL WOUND SURGICAL DEBRIDEMENT (Cardiac disorders) | 1 (1) | 0 (0)
URINARY TRACT INFECTION, HYPERGLYCEMIA (Infections and infestations) | 0 (0) | 1 (1)
UTI WITH SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Eflornithine and Sulindac) (N=191) | Arm II (Placebo) (N=184)
5 LBS X 2 WKS (Investigations) | 0 (0) | 1 (1)
A-FIB (Cardiac disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 (6) | 5 (5)
ABDOMINAL PAIN ABD CRAMPING AND BLOAT (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN ABD. CRAMP AND CONSTIPATION (Gastrointestinal disorders) | 1 (2) | 0 (0)
ABDOMINAL PAIN ABDOMINAL CRAMPING (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN CRAMPING (Gastrointestinal disorders) | 2 (2) | 0 (0)
ABDOMINAL PAIN CRAMPS/ CONSTIPATION (Gastrointestinal disorders) | 1 (2) | 0 (0)
ABDOMINAL PAIN DIARRHEA X 1-2 DAILY, CRAMPING (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN DIARRHEA X 3-4 DAILY, CRAMPING (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN EPIGASTRIC PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN LEFT SIDE (Gastrointestinal disorders) | 2 (2) | 0 (0)
ABDOMINAL PAIN LOWER ABDOMEN, INTERMITTENT (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN LOWER ABDOMINAL CRAMPING AFTER COLONOSCOPY (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN OCCASIONAL ABD CRAMP WITH LOOSE STOOL WHEN NERVIOUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN STOMACH CRAMPS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPSET STOMACH (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABNORMAL PSA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ABNORMAL X-RAY (Investigations) | 1 (1) | 0 (0)
ANKLE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 8 (9) | 3 (6)
ANOREXIA DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ANOREXIA LOSS OF APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 4 (4)
ANXIETY AND DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
ANXIETY DEPRESSION (Psychiatric disorders) | 1 (2) | 0 (0)
ANXIETY INCREASED ANXIERTY AND BOREDOM (Psychiatric disorders) | 0 (0) | 1 (1)
ANXIETY MOOD SWINGS, HOT FLASHES, ANXIETY (Psychiatric disorders) | 1 (3) | 0 (0)
APPETITE LOSS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHIALGIA SHOULDER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ARTHRITIS ARTHRITIS FLARE UP - HANDS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ARTHRITIS BACK PAIN WORSENING (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ARTHRITIS BILATERAL KNEE PAIN R/T (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ARTHRITIS EXACERBATION OF GOUT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ARTHRITIS GOUT, RIGHT FOOT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ARTHRITIS HAND PAIN (ARTHRITIS) OR (FIBROMYALGIA EPISODE) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ARTHRITIS IN RIGHT KNEE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ARTHRITIS LEFT HAND JOINT PAIN R/T ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ARTHRITIS LEFT KNEE/ LEFT WRIST (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
ARTHRITIS LEFT WRIST (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
ARTHRITIS NECK (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ARTHRITIS OSTEO (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ARTHRITIS OSTEOARTHRITIS-LEFT KNEE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ARTHRITIS OSTEOARTHRITIS-LEFT WRIST (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ARTHRITIS R THUMB JOINT PAIN R/T (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ARTHRITIS RIGHT ELBOW (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ARTHRITIS THUMB PAIN - ARTHRITIS BOTH HANDS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ARTHRITIS TOE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ASTHMA FLARE-UP (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
BACK PAIN (MOTRIN USE) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BACK PAIN, ON MOTRIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BACK STRAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BALANCE (Nervous system disorders) | 4 (4) | 3 (3)
BALANCE BALANCE DISTURBANCE (Nervous system disorders) | 2 (2) | 1 (2)
BALANCE BALANCE DISTURBANCE DUE TO B12 MALABSORPTION (Nervous system disorders) | 0 (0) | 1 (1)
BALANCE DISTANCE DISTURBANCE (Nervous system disorders) | 1 (1) | 0 (0)
BALANCE DISTURBANCE (Nervous system disorders) | 4 (4) | 0 (0)
BASAL CELL SKIN LESION REMOVAL (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
BASAL CELL TAKEN FROM FACE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
BELLS PALSY SIDE WEAKNESS (Nervous system disorders) | 1 (1) | 0 (0)
BIL LE EDEMA (General disorders) | 1 (1) | 0 (0)
BIL SWOLLEN FEET AND ANKLES (General disorders) | 1 (1) | 0 (0)
BIL. CATARACTS (Eye disorders) | 0 (0) | 1 (1)
BLACK STOOLS (THINKS FROM MAALOX) (Gastrointestinal disorders) | 1 (1) | 0 (0)
BLEEDING GUMS DURING DENTAL VISIT (Gastrointestinal disorders) | 0 (0) | 2 (2)
BLEEDING IN EYE FROM THORN (Eye disorders) | 1 (1) | 0 (0)
BLEEDING RECTAL (Gastrointestinal disorders) | 7 (12) | 5 (6)
BLEEDING RECTAL 4 EPISODES BRBPR (Gastrointestinal disorders) | 1 (1) | 0 (0)
BLEEDING RECTAL BRB TOILET PAPER (Gastrointestinal disorders) | 0 (0) | 1 (2)
BLEEDING RECTAL HEMORRHOIDS (Gastrointestinal disorders) | 5 (5) | 2 (2)
BLEEDING* BLOOD IN THE URINE (Renal and urinary disorders) | 0 (0) | 1 (1)
BLEEDING* BLOOD IN URINE (Renal and urinary disorders) | 0 (0) | 3 (3)
BLEEDING* EAR CANALS, LEFT AND RIGHT (Ear and labyrinth disorders) | 0 (0) | 1 (1)
BLEEDING* EPITAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BLEEDING* GUMS (Infections and infestations) | 0 (0) | 1 (1)
BLEEDING* HEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
BLEEDING* HEMATURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
BLEEDING* HEMATURIA - TRACE (Renal and urinary disorders) | 0 (0) | 1 (1)
BLEEDING* HEMORRHAGE HEMATURIA (Renal and urinary disorders) | 1 (2) | 0 (0)
BLEEDING* NOSE BLEED (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
BLEEDING* PENILE (Reproductive system and breast disorders) | 0 (0) | 1 (3)
BLEEDING* PROLONGED MENSTRUAL BLEEDING (Reproductive system and breast disorders) | 1 (1) | 0 (0)
BLEEDING* SHAVING (General disorders) | 0 (0) | 1 (1)
BLEEDING* UPPER GI BLEED (Gastrointestinal disorders) | 0 (0) | 1 (1)
BLEEDING* VAGINAL (Reproductive system and breast disorders) | 0 (0) | 1 (1)
BLEEDING* VAGINAL BLEED (Reproductive system and breast disorders) | 1 (2) | 0 (0)
BLEEDING, RECTAL (Gastrointestinal disorders) | 2 (2) | 0 (0)
BLOOD IN STOOL (Gastrointestinal disorders) | 4 (4) | 0 (0)
BLOOD IN STOOL /HEMORRHOID (Gastrointestinal disorders) | 1 (1) | 0 (0)
BLOOD IN STOOL BURGUNDY (Gastrointestinal disorders) | 1 (1) | 0 (0)
BLOOD IN STOOL DIARRHEA, CRAMPING, BLACK STOOL (Gastrointestinal disorders) | 0 (0) | 1 (1)
BLOOD IN STOOL DX: COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
BLOOD IN STOOL OCCULT (Gastrointestinal disorders) | 1 (1) | 0 (0)
BLOOD IN STOOL SMALL DOT (Cardiac disorders) | 1 (1) | 0 (0)
BLOOD IN URINE (Renal and urinary disorders) | 0 (0) | 1 (2)
BLOOD WITH BM (Gastrointestinal disorders) | 0 (0) | 1 (1)
BOWEL MOVEMENT REGULARITY CONTINUES (Gastrointestinal disorders) | 0 (0) | 1 (1)
BPH (Reproductive system and breast disorders) | 1 (1) | 0 (0)
BROKE BACK (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BROKEN ANKLE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BROKEN TOE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BROKEN TOOTH (Infections and infestations) | 1 (1) | 0 (0)
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BRUISING LEFT HIP AREA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
BX - BPH (Reproductive system and breast disorders) | 0 (0) | 1 (1)
CAD (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC* ALTERED LEFT VENTRICULAR DIASTOLIC FUNCTION (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC* ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 2 (2)
CARDIAC* CONGESTIVE HEART FAILURE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC* DX -- POSSIBLE RETURN OF RENOVASCULAR HTN (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC* DX WITH CAD (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC* FLUID IN LUNGS (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC* HEART ATTACK (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC* HEART MURMUR (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC* HEART PALPITATIONS AND HYPERTENSION (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC* LEFT BUNDLE BRANCH BLOCK (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC* MILD AORTIC SCLEROSIS (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC* MYOCARDIAL INFARCTION BY EKG (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC* NEAR FAINT EPISODES, DX HTN, ON DRUGS (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC* PALPITATION (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC* PALPITATIONS (PSVT) (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC* TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC* TACHYCARDIA EPISODES - INCREASED FREQUENCY (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC* UNSTABLE ANGINA, CHEST PAIN (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC* VALVULAR HEART DISEASE - MILVAL VALVE REGURGITATION (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC* VASOVAGAL EPISODE (Cardiac disorders) | 1 (2) | 0 (0)
CARDIAC* VASOVAGAL SYNCOPAL EPISODE (Cardiac disorders) | 0 (0) | 1 (1)
CARPAL TUNNEL SYNDROM (Nervous system disorders) | 0 (0) | 1 (1)
CATARACT SURGERY RIGHT EYE (Eye disorders) | 0 (0) | 1 (1)
CELLULITIS - LEFT BREAST WOUND - NON INFECTIOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
CELLULITIS LEF SIDE FACE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
CENTRAL NERVOUS SYSTEM (Nervous system disorders) | 1 (1) | 0 (0)
CENTRAL NERVOUS SYSTEM DEPRESSION (Nervous system disorders) | 0 (0) | 1 (1)
CENTRAL NERVOUS SYSTEM HEADACHE RELATED TO CHOCOLATE (Nervous system disorders) | 1 (1) | 0 (0)
CENTRAL NERVOUS SYSTEM INCREASE IN SEIZURES (Nervous system disorders) | 1 (1) | 0 (0)
CENTRAL NERVOUS SYSTEM MEMORY LOSS (Nervous system disorders) | 0 (0) | 1 (1)
CENTRAL NERVOUS SYSTEM MEMORY LOSS INCREASED (Nervous system disorders) | 1 (1) | 0 (0)
CENTRAL NERVOUS SYSTEM MEMORY LOSS/FORGETFULNESS (Nervous system disorders) | 0 (0) | 1 (1)
CENTRAL NERVOUS SYSTEM MEMORY PROBLEMS (Nervous system disorders) | 1 (1) | 0 (0)
CHANGE (Ear and labyrinth disorders) | 1 (1) | 0 (0)
CHANGE IN HEARING PER AUDIOGRAM (Ear and labyrinth disorders) | 1 (1) | 0 (0)
CHANGE IN SIGNIFICANT OTHER'S PERCEPTION OF HEARING (Ear and labyrinth disorders) | 1 (1) | 0 (0)
CHEST PAIN RELATED TO 4/18 REPORT FOR HEART BURN (Cardiac disorders) | 1 (1) | 0 (0)
CHEST PAIN WITH EXERTION (Cardiac disorders) | 1 (1) | 0 (0)
CN VIII (Ear and labyrinth disorders) | 0 (0) | 1 (1)
COLD (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
COLD SYMPTOMS (General disorders) | 11 (13) | 9 (11)
COLD SYMPTOMS COLD X3-4 (General disorders) | 1 (1) | 0 (0)
COLD SYMPTOMS COUGH AND COLD SYMPTOMS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COLD SYMPTOMS DX SINUS INFECTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COLD SYMPTOMS HEAD (General disorders) | 1 (1) | 0 (0)
COLD SYMPTOMS HEAD COLD (General disorders) | 0 (0) | 6 (6)
COLD SYMPTOMS NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COLD SYMPTOMS POST NASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COLD SYMPTOMS SINUS DRAINAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COLD SYMPTOMS SNIFFLES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COLD SYMPTOMS SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COLD SYMPTOMS WITH COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COLD WITH URI SX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COLD/SINUS/EAR CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 6 (8) | 4 (7)
CONSTIPATION CHRONIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONSTIPATION GETTING WORSE (Gastrointestinal disorders) | 1 (1) | 0 (0)
CONSTIPATION INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONSTIPATION R/T IMMODIUM (Gastrointestinal disorders) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COUGH* (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 5 (8)
COUGH* DRY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CRAMPING (Gastrointestinal disorders) | 1 (1) | 0 (0)
CUT SHIN = INFECTION (CELLULITIS) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CYST. DERMAL ON BACK (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
DECREASE HGB 5% FROM BASELINE (Investigations) | 0 (0) | 1 (1)
DECREASE IN HGB (Investigations) | 0 (0) | 1 (1)
DECREASED PERIPHERAL REFLEXES (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 2 (5)
DEPRESSION, MOM'S DEATH (Psychiatric disorders) | 1 (1) | 0 (0)
DERMATOLOGY* 2 SPOTS ON SCALP (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOLOGY* ACTINIC KERATOSES REMOVED X3 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOLOGY* ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOLOGY* ANAL SKIN TAG REMOVED (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOLOGY* BASAL CELL CARCINOMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOLOGY* BCC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOLOGY* BLACK SPOT CHANGES ON SCALP (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY* BOIL (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
DERMATOLOGY* BRUISES (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY* BRUISING INTERMITTENT (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY* DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY* DERMATITIS/ EXACERBATION THUMBS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOLOGY* DISCOVERY AND REMOVAL OF BENIGN SKIN LESION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY* DRY SKIN, FEET (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOLOGY* EXTREME RASH ON TRUNK (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY* FACIAL EDEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOLOGY* FUNGAL INF. (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOLOGY* IMPETIGO (NOSE) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOLOGY* MELANOMA UPPER ARM MOLE SKIN EXCISION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOLOGY* PERIANA PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY* PIGMENTATION SLOW TO FILL IN ON SCRAPE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY* PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
DERMATOLOGY* R/O POSSIBLE SKIN CA SPOT SCHAGE COLOR AND SIZE, BX 2/12/04 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY* RASH RIGHT ARM (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY* REMOVAL SKIN CA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY* ROSACEA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
DERMATOLOGY* ROSACEA FLARE-UP (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY* SKIN - BUMP, RED LEFT UPPER MOUTH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOLOGY* SKIN - LESION RIGHT EAR ANTIHELIX (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY* SKIN LESION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY* SKIN LESION ABOVE FOREHEAD (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY* SKIN LESIONS (REMOVED) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY* SKIN RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
DERMATOLOGY* SKIN ROSACEA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY* SKIN SENSITIVE TO SUN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DIABETES NEW ONSET (Endocrine disorders) | 0 (0) | 1 (1)
DIAPHORESIS ABDOMINAL DISCOMFORT (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 31 (49) | 29 (47)
DIARRHEA + ABDOMINAL CRAMPS (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHEA 2 EPISODES (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHEA 3 EPISODES (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHEA AFTER COLONOSCOPY (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHEA CONTINUED DIARRHEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHEA LOOSE STOOL (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHEA LOOSER STOOL (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHEA MILD (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHEA OCCASIONAL (Gastrointestinal disorders) | 1 (1) | 1 (1)
DIARRHEA X 1 RELATED TO FOOD (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIVERTICULITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 8 (11) | 8 (11)
DIZZINESS AFT CERUMEN REMOVAL (Nervous system disorders) | 0 (0) | 1 (1)
DIZZINESS FELL R/T LIGHT HEADED (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS VERTIGO (Nervous system disorders) | 0 (0) | 1 (1)
DIZZINESS/VERTIGO (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS/VERTIGO EPISODE LASTING LESS THAN 10 SEC (Nervous system disorders) | 1 (1) | 0 (0)
DROP HGB (Investigations) | 0 (0) | 1 (1)
DROP IN HGB (Investigations) | 0 (0) | 1 (1)
DRY EYE (Eye disorders) | 0 (0) | 1 (1)
DX CHF (Cardiac disorders) | 0 (0) | 1 (1)
DX WITH EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNEA ON EXERTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
EAR INFECTION (Ear and labyrinth disorders) | 1 (1) | 2 (2)
EARLY SATIETY (Gastrointestinal disorders) | 0 (0) | 1 (1)
ELECT. BALANCE (Investigations) | 1 (1) | 0 (0)
ELEVATED BLOOD PRESSURE (Cardiac disorders) | 1 (1) | 0 (0)
ELEVATED CREATININE BUN (Investigations) | 1 (2) | 0 (0)
ELEVATED LIVER ENZYMES (Investigations) | 0 (0) | 1 (1)
ELEVATED PSA (Investigations) | 0 (0) | 1 (1)
ELEVATED TRIGLYCERIDE (Investigations) | 0 (0) | 1 (1)
ELEVATED TRIGLYCERIDES 571 (Investigations) | 0 (0) | 1 (1)
ELEVATED TRIGLYCERIDES 779 (Investigations) | 0 (0) | 1 (1)
ENLARGED THYROID (Endocrine disorders) | 1 (1) | 0 (0)
EPIGASTRIC PAIN (Gastrointestinal disorders) | 8 (8) | 7 (8)
EPIGASTRIC PAIN 2-3 EPISODES PER WEEK (Gastrointestinal disorders) | 0 (0) | 1 (1)
EPIGASTRIC PAIN GAS PAINS (Gastrointestinal disorders) | 0 (0) | 1 (1)
EPIGASTRIC PAIN GAS X 1 PER MONTH (Gastrointestinal disorders) | 0 (0) | 1 (1)
EPIGASTRIC PAIN GASTRIC PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
EPIGASTRIC PAIN GERD (Gastrointestinal disorders) | 1 (1) | 1 (1)
EPIGASTRIC PAIN GERD (INCREASE SYMPTOMS) (Gastrointestinal disorders) | 0 (0) | 1 (1)
EPIGASTRIC PAIN GERD, WORSENED, EST. START 1970 (Gastrointestinal disorders) | 0 (0) | 1 (1)
EPIGASTRIC PAIN PAIN X 1 (Gastrointestinal disorders) | 0 (0) | 1 (1)
EPIGASTRIC PAIN RIGHT SIDE (Gastrointestinal disorders) | 0 (0) | 1 (1)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ERECTILE DYSFUNTION (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ERYTHORMATOUS PLAQUES (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
EXACERBATION OF LEFT KNEE PAIN - ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
EXCISED MASS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 32 (34) | 17 (19)
FATIGUE* ALLERGY FATIGUE (General disorders) | 0 (0) | 1 (1)
FATIGUE* BILATERAL LEG FATIGUE (General disorders) | 0 (0) | 1 (1)
FATIGUE* DIAPHORESIS AFTER MEALS (General disorders) | 0 (0) | 1 (1)
FATIGUE* INCREASED (General disorders) | 0 (0) | 1 (1)
FATIGUE* MILD (General disorders) | 0 (0) | 1 (1)
FATIGUE* MILD DEPRESSION (General disorders) | 0 (0) | 1 (1)
FATIGUE* MUSCLE ACHES (General disorders) | 0 (0) | 1 (1)
FATIGUE* POSSIBLE VIRUS (General disorders) | 0 (0) | 1 (1)
FATIGUE* R/T MUSCLE WEAKNESS (General disorders) | 0 (0) | 1 (1)
FATIGUE* RELATED TO MUSCLE WEAKNESS (General disorders) | 0 (0) | 1 (1)
FATIGUE* SYNCOPE (General disorders) | 1 (1) | 0 (0)
FATIGUE* WEAKNESS (General disorders) | 1 (1) | 0 (0)
FEELING HEATED AFTER TAKING MEDICATION (Psychiatric disorders) | 1 (1) | 0 (0)
FEVER (General disorders) | 2 (2) | 1 (1)
FEVER BLISTERS (Infections and infestations) | 0 (0) | 1 (1)
FEVER INTERMITTENT (General disorders) | 1 (1) | 0 (0)
FEVER SWEATS (General disorders) | 0 (0) | 1 (2)
FEVER X 2DAYS (General disorders) | 1 (1) | 0 (0)
FEVER X1 (General disorders) | 1 (1) | 0 (0)
FINGER LACERATION RIGHT HAND (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (1)
FLU (General disorders) | 7 (7) | 3 (3)
FLU ACHY, NAUSEA, HEADACHE, COUGH (General disorders) | 1 (1) | 0 (0)
FLU DIARRHEA N/V (General disorders) | 1 (2) | 0 (0)
FLU FLU-LIKE SYMPTOMS (General disorders) | 1 (1) | 0 (0)
FLU INFECTION (General disorders) | 1 (1) | 0 (0)
FLU S/S (General disorders) | 0 (0) | 1 (1)
FLU SYMPTOMS (General disorders) | 1 (1) | 1 (1)
FLU X5 DAYS (General disorders) | 1 (1) | 0 (0)
FLU-LIKE SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
FOOT CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FORHEAD LESION REMOVAL (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
FUZZY EYESIGHT (Eye disorders) | 0 (0) | 1 (1)
FX RT GREAT TOE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
GASTRIC REFLUX (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GENITOURINARY - URINATING (Renal and urinary disorders) | 1 (1) | 0 (0)
GENITOURINARY URINATING (Renal and urinary disorders) | 1 (1) | 0 (0)
GI ABDOMINAL BLOATING (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI BARRETT'S ESOPHAGUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI BARRETT'S ESOPHAGUS/DYSPLASIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI BLOATING (Gastrointestinal disorders) | 2 (2) | 0 (0)
GI BLOATING / GAS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI BLOATING/FEELING OF INCOMPLETE EVACUATION, CONSISTENT WITH IBS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI CECUM BIOPSY: EROSIM WITH CHRONIC INFLAMMATION, NON-SPECIFIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI CONT. COLITIS SX (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI CONT. ESOPHAGEAL IRRITATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI ESOPHAGEAL FULLNESS RELATED TO GASTRO CIRCLAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI HEARTBURN (Gastrointestinal disorders) | 1 (1) | 3 (3)
GI HEARTBURN 1 - 2 EPISODES/WEEK (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI HEARTBURN 4 EPISODES WEEKLY (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI HEARTBURN 5-6 EPISODES/WEEK (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI HEARTBURN 5-6- EPISODES/WEEK (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI HEARTBURN X9 EPISODES (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI HEARTBURN, 1 EPISODE PER WEEK (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI INCREASE IN GERD SYMPTOMS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI INCREASED GERD SX (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI INFLAMMATION COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI PEPTIC ULCER DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI STOMACH CRAMPS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI UPPER GI PAIN/ACID REFLUX (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI UPSET (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI UPSET STOMACH (Gastrointestinal disorders) | 0 (0) | 2 (3)
GI UPSET STOMACH X 2 EPISODES (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI UPSET STOMACH X3 EPISODES (Gastrointestinal disorders) | 1 (1) | 0 (0)
GLUCOSURIA (Renal and urinary disorders) | 2 (2) | 0 (0)
GOUT (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
GROIN PULL (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
GUM SORENESS (Gastrointestinal disorders) | 0 (0) | 1 (2)
H. PYLORI +, STOMACH UPSET (Gastrointestinal disorders) | 1 (1) | 0 (0)
H.PYLORI +, DX IBS - CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAND PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HAND SURGERY - TRIGGER FINGER (Surgical and medical procedures) | 1 (1) | 0 (0)
HEAD CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 19 (22) | 18 (26)
HEADACHE INTERMITTENT (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE NAUSEA (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE PAIN 5 EPISODES (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE PRESSURE (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE SIDE (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE SINUS PAIN (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE WITH NAUSEA AND VOMITING (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE WITH NAUSEA AND VOMITTING (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE WITH VISION INVOLVEMENT (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE X1 (Nervous system disorders) | 0 (0) | 1 (1)
HEARING (Ear and labyrinth disorders) | 5 (5) | 5 (7)
HEARING "CARBONIZATION SOUND" - LEFT EAR (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING /INNER EAR - "STATIC NOISE" LEFT (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING AUDIO CHANGE (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING AUDIO CHANGE SUBCLINICAL (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING AUDIO SHOWS NO CHANGE (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING AUDIOGRAM (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING AUDIOGRAM CHANGE (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING AUDIOGRAM GRADE 1 HEARING CHANGE (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING AUDIOGRAM ONLY (Ear and labyrinth disorders) | 2 (2) | 0 (0)
HEARING AUDIOMETIC CHANGE, OFF STUDY (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING AUDIOMETRIC CHANGE (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING AUDIOMETRIC CHANGE BILATERAL (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING AUDIOMETRIC CHANGE LEFT EAR (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING AUDIOMETRIC CHANGE RIGHT EAR (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING AUDIOMETRIC CHANGE RIGHT EAR/ OVERALL NO SIGNIFICANT CHANGE (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING AUDITORY (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING CHANGE (Ear and labyrinth disorders) | 11 (13) | 6 (6)
HEARING CHANGE AUDIOGRAM (Ear and labyrinth disorders) | 2 (2) | 1 (1)
HEARING CHANGE NOTED ON AUDIO (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING CHANGE PER AUDIOGRAM (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING CHANGE-LEFT EAR (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING CHANGE? PT NOT SURE (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING DECREASE IN HEARING (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING DECREASE IN HEARING ABILITY (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING DECREASE LEFT>RIGHT (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING DECREASED (Ear and labyrinth disorders) | 1 (1) | 1 (1)
HEARING DECREASED RIGHT EAR (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING DIFFICULTY (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING HEARING CHANGE (Ear and labyrinth disorders) | 3 (3) | 3 (3)
HEARING HEARING LOSS (Ear and labyrinth disorders) | 2 (2) | 3 (3)
HEARING HEARING LOSS - SIGNIFICANT OTHER PERCEPTION (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING HEARING LOSS AUDIOMETRY ONLY (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING HEARNING LOSS/ SUBCLINICAL (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING HEARS PULSE IN LEFT EAR (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING HUSBAND THINKS POSSIBLE HEARING CHANGE (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING INNER EAR (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING LOSS (Ear and labyrinth disorders) | 3 (3) | 2 (3)
HEARING LOSS (SELF-PERCEPTION) (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING LOSS + PAIN, LEFT NECK (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING LOSS - SIGNIFICANT OTHER PERCEPTION (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING LOSS IN LEFT EAR (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING LOSS IN LEFT EAR, AUDIO DONE 11-30-00 (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING MILD LOSS (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING MUFFLED (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING OTITIS MEDIA (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING OTOTOXICITY (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING OTOTOXICITY - AUDIOGRAM ONLY (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING PLUGGED RIGHT EAR (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING POSSIBLE CHANGE (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING RIGHT EAR "PLUGGED" X2 EPISODES (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING RIGHT EAR PAIN/PLUG (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING RIGHT EAR PAIN/PLUG, EUSTACHIAN TUBE DYSFUNCTION (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEARING SELF PERCEPTION (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING SELF PERCEPTION, DIFFICULTY WITH DISCRIMINATION (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING SLIGHT LOSS (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HEARING TINNITUS (HAS GOTTEN SLIGHTLY WORSE OVER LAST 2 MONTHS) (Ear and labyrinth disorders) | 0 (0) | 1 (1)
HEART DISEASE (Cardiac disorders) | 0 (0) | 1 (1)
HEARTBURN (Gastrointestinal disorders) | 1 (1) | 1 (2)
HEMATARIA (Renal and urinary disorders) | 1 (1) | 0 (0)
HEMATURIA-MICROSCOPIC (Renal and urinary disorders) | 1 (1) | 0 (0)
HEMIANOPSIA (Eye disorders) | 0 (0) | 1 (1)
HEMMORRHOID (Gastrointestinal disorders) | 1 (1) | 0 (0)
HEMOGLOBINURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
HEMORRHOIDS (Gastrointestinal disorders) | 2 (2) | 3 (4)
HEMORRHOIDS FLARE-UP (Gastrointestinal disorders) | 0 (0) | 1 (1)
HERNIA REPAIR (Surgical and medical procedures) | 0 (0) | 1 (1)
HERPES (Infections and infestations) | 1 (1) | 0 (0)
HIGH BLOOD PRESSURE (Cardiac disorders) | 1 (1) | 0 (0)
HIP AREA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HIP BURSITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HIP PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
HOT FLASHES (Vascular disorders) | 1 (1) | 0 (0)
HTN (Cardiac disorders) | 1 (1) | 0 (0)
HYPERGLICEMIA (Investigations) | 1 (2) | 0 (0)
HYPERGLYCEMIA (Investigations) | 1 (1) | 2 (2)
HYPERKALEMIA (Investigations) | 2 (2) | 0 (0)
HYPERTENSION (Cardiac disorders) | 6 (7) | 6 (7)
HYPERTENSION /DIABETES (Cardiac disorders) | 1 (1) | 0 (0)
HYPERTENSION MILD/MOD (Cardiac disorders) | 1 (1) | 0 (0)
HYPERTENSION RETURNED (Cardiac disorders) | 1 (1) | 0 (0)
HYPERTENSION SUSPECT OCULAR HYPERTENSION (Cardiac disorders) | 1 (1) | 0 (0)
HYPERTENSION UNCONTROLLED (Cardiac disorders) | 0 (0) | 1 (1)
INCREASE "BURPING" (Gastrointestinal disorders) | 1 (1) | 0 (0)
INCREASE BP WITH RINGING IN EARS (Cardiac disorders) | 0 (0) | 1 (1)
INCREASE FLATULENCE (Gastrointestinal disorders) | 1 (1) | 0 (0)
INCREASE FREQ OF HEMORHOIDAL BLEEDING (Gastrointestinal disorders) | 1 (1) | 0 (0)
INCREASE STOOL FREQUENCY (Gastrointestinal disorders) | 1 (1) | 0 (0)
INCREASE STOOLING (Gastrointestinal disorders) | 1 (1) | 0 (0)
INCREASED ALKPHOSPHATASE (Investigations) | 1 (1) | 0 (0)
INCREASED ALT (Investigations) | 1 (1) | 0 (0)
INCREASED AST (Investigations) | 1 (1) | 0 (0)
INCREASED BILIRUBIN (Investigations) | 1 (1) | 0 (0)
INCREASED BOWEL MOVEMENTS (Gastrointestinal disorders) | 0 (0) | 1 (1)
INCREASED CREATININE (Investigations) | 1 (1) | 0 (0)
INCREASED FATIGUE (General disorders) | 0 (0) | 1 (1)
INCREASED FLATULENCE; ANAL INCONTINENCE (Gastrointestinal disorders) | 1 (2) | 0 (0)
INCREASED FREQUENCY OF DROPPING ITEMS (Nervous system disorders) | 1 (1) | 0 (0)
INCREASED HEMOGLOBIN (Investigations) | 0 (0) | 1 (1)
INCREASED LFTS (Investigations) | 0 (0) | 1 (1)
INCREASED ORAL HERPES OUTBREAKS (Infections and infestations) | 0 (0) | 1 (1)
INCREASED STOOLING (Gastrointestinal disorders) | 0 (0) | 1 (1)
INDIGESTION (Gastrointestinal disorders) | 4 (6) | 3 (3)
INDIGESTION DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
INDIGESTION EPIGASTRIC PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
INDIGESTION HEART BURN (Gastrointestinal disorders) | 1 (1) | 0 (0)
INFECTION* BLADDER (Infections and infestations) | 0 (0) | 2 (2)
INFECTION* BLADDER INFECTION (Infections and infestations) | 1 (1) | 0 (0)
INFECTION* EAR (Infections and infestations) | 0 (0) | 2 (2)
INFECTION* ESOPHAGITIS (Infections and infestations) | 1 (1) | 0 (0)
INFECTION* EUSTACHIAN TUBES (Infections and infestations) | 1 (1) | 0 (0)
INFECTION* FUNGAL FINGERNAIL (Infections and infestations) | 1 (1) | 0 (0)
INFECTION* FUNGAL INFECTION FINGERNAILS (Infections and infestations) | 1 (1) | 0 (0)
INFECTION* FUNGAL, LEFT MIDDLE FINGER (Infections and infestations) | 1 (1) | 0 (0)
INFECTION* INFECTED SCROTAL CYST (Infections and infestations) | 1 (1) | 0 (0)
INFECTION* INSECT BITE RIGHT ANKLE (Infections and infestations) | 1 (1) | 0 (0)
INFECTION* LEFT INDEX FINGER (Infections and infestations) | 1 (1) | 0 (0)
INFECTION* LEFT LOWER LEG AK SITE (Infections and infestations) | 1 (1) | 0 (0)
INFECTION* LEFT TESTICLE (Infections and infestations) | 0 (0) | 1 (1)
INFECTION* MIDDLE EAR-BLOCKED EUSTACHIAN TUBE (Infections and infestations) | 1 (1) | 0 (0)
INFECTION* PNEUMONIA POSS "SCAR" ON CXR (Infections and infestations) | 1 (1) | 0 (0)
INFECTION* RIGHT BREAST (Infections and infestations) | 0 (0) | 1 (1)
INFECTION* RIGHT CALF BITE (Infections and infestations) | 0 (0) | 1 (2)
INFECTION* RIGHT MIDDLE FINGER NAIL (Infections and infestations) | 1 (1) | 0 (0)
INFECTION* SINUS (Infections and infestations) | 3 (4) | 0 (0)
INFECTION* SINUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
INFECTION* SKIN FUNGAL (Infections and infestations) | 0 (0) | 1 (1)
INFECTION* TOOTH (Infections and infestations) | 2 (2) | 1 (2)
INFECTION* UPPER RESPIRATORY (Infections and infestations) | 0 (0) | 1 (1)
INFECTION* VAGINAL YEAST (Infections and infestations) | 1 (1) | 1 (1)
INFECTION* WOUND/INFECTION LEFT LE (Infections and infestations) | 0 (0) | 1 (1)
INFECTION* YEAST (Infections and infestations) | 1 (1) | 0 (0)
IRRITABILITY (Psychiatric disorders) | 0 (0) | 1 (1)
ITCHING AND RASH TO RECTUM (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
JOINT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
JOINT PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
KIDNEY PROBLEMS (Renal and urinary disorders) | 1 (1) | 0 (0)
KIDNEY PROBLEMS/RENAL-OTHER (Renal and urinary disorders) | 1 (1) | 0 (0)
KIDNEY STONE (Renal and urinary disorders) | 0 (0) | 1 (1)
KIDNEY STONES (Renal and urinary disorders) | 1 (1) | 0 (0)
KNEE PAIN (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
LABS 10 % HGB DROP (Investigations) | 0 (0) | 1 (1)
LABS 10% DROP HGB (Investigations) | 1 (1) | 0 (0)
LABS 10% DROP HGB WITH DYSMENORRHEA (Investigations) | 0 (0) | 1 (1)
LABS 10% DROP IN HGB (Investigations) | 0 (0) | 1 (1)
LABS ANEMIA (Investigations) | 2 (2) | 0 (0)
LABS ANEMIA - DROP IN HGB (Investigations) | 0 (0) | 1 (2)
LABS ANEMIA, MENSUS DISORDER (Investigations) | 0 (0) | 1 (1)
LABS ANEMIA: IRON DEFICIENCY (Investigations) | 1 (1) | 0 (0)
LABS B-12 DEFICIENCY (Investigations) | 1 (1) | 1 (1)
LABS BLOOD GLUCOSE ELEVATED (Investigations) | 0 (0) | 1 (2)
LABS DECREASE HGB GREATER THAN 10% (Investigations) | 1 (1) | 0 (0)
LABS DECREASE IN HGB (Investigations) | 4 (4) | 4 (4)
LABS DECREASED HBG 10% FROM BASELINE (Investigations) | 1 (1) | 0 (0)
LABS DECREASED HBG OF 10% BASELINE (Investigations) | 1 (1) | 0 (0)
LABS DECREASED HEMOGLOBIN (Investigations) | 0 (0) | 2 (2)
LABS DECREASED HEMOGLOBIN >10% (Investigations) | 0 (0) | 1 (1)
LABS DECREASED HEMOGLOBIN NOT GREATER THAN 10% BASELINE (Investigations) | 1 (1) | 0 (0)
LABS DECREASED HEMOGLOBIN, REDRAW 12/4/01 (Investigations) | 1 (1) | 0 (0)
LABS DECREASED HGB (Investigations) | 1 (1) | 1 (1)
LABS DECREASED HGB GREATER THAN 10% BASELINE (Investigations) | 1 (1) | 0 (0)
LABS DECREASED HGB GREATER THAN 10% FROM BASELINE (Investigations) | 1 (1) | 0 (0)
LABS DECREASED HGB, 10% FROM BASELINE (Investigations) | 1 (1) | 0 (0)
LABS DECREASED HGB: CHRONIC (Investigations) | 1 (1) | 0 (0)
LABS DECREASED NEUTROPHILS (Investigations) | 0 (0) | 1 (1)
LABS DECREASED WBC (Investigations) | 4 (4) | 0 (0)
LABS DROP IN HGB AND HEMATOCRIT (Investigations) | 1 (1) | 0 (0)
LABS ELEVATED ALKALINE PHOSPHATASE (Investigations) | 0 (0) | 1 (1)
LABS ELEVATED BILIRUBIN (Investigations) | 1 (1) | 0 (0)
LABS ELEVATED PSA (Investigations) | 1 (1) | 2 (2)
LABS ENDOCRINE: ELEVATED BLOOD GLUCOSE (Investigations) | 1 (1) | 0 (0)
LABS HEMATURIA (Investigations) | 3 (3) | 0 (0)
LABS HGB DECREASE = 10% (Investigations) | 1 (1) | 0 (0)
LABS HGB DECREASE GREATER THAN 10% (Investigations) | 1 (1) | 0 (0)
LABS HGB DROP 10% (Investigations) | 1 (2) | 0 (0)
LABS HIGH ALT (Investigations) | 0 (0) | 1 (1)
LABS HIGH AST (Investigations) | 0 (0) | 1 (1)
LABS HIGH CHOLESTEROL LEVELS (Investigations) | 0 (0) | 1 (1)
LABS HYPERCHOLESTEREMIA (Investigations) | 0 (0) | 1 (1)
LABS HYPERKALEMIA (Investigations) | 0 (0) | 1 (1)
LABS HYPERLIPIDEMIA (Investigations) | 3 (3) | 0 (0)
LABS INCREASED ALKALINE PHOSPHATASE (Investigations) | 0 (0) | 1 (1)
LABS INCREASED CHOLESTEROL (Investigations) | 1 (1) | 0 (0)
LABS INCREASED GLUCOSE (Investigations) | 0 (0) | 1 (1)
LABS INCREASED HGB A1C (Investigations) | 0 (0) | 1 (1)
LABS LOW BLOOD SUGAR (Investigations) | 0 (0) | 1 (1)
LABS LOW HEMOGLOBIN (Investigations) | 0 (0) | 1 (1)
LABS LOW HEMOGLOBIN AFTER SURGERY (Investigations) | 1 (1) | 0 (0)
LABS LOW HGB (Investigations) | 1 (1) | 0 (0)
LABS LOW HGB - 10% FROM BASELINE (Investigations) | 0 (0) | 3 (3)
LABS LOW HGB = 10% (Investigations) | 1 (1) | 0 (0)
LABS LOWER WBC (Investigations) | 0 (0) | 1 (1)
LABS PROTEINURIA (Investigations) | 1 (5) | 0 (0)
LABS PSA ELEVATION (Investigations) | 1 (1) | 0 (0)
LABS PSA LEVELS INCREASED (5 TO 8 TO 11) (Investigations) | 1 (1) | 0 (0)
LABS WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 (0) | 1 (1)
LABS WHITE BLOOD CELLS COUNT DOWN (Investigations) | 1 (1) | 0 (0)
LEFT EAR INFECTION, RINGING WITH FULLNESS (Ear and labyrinth disorders) | 0 (0) | 1 (1)
LEFT FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LEFT KIDNEY STONE (Renal and urinary disorders) | 0 (0) | 1 (1)
LEFT KNEE (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
LEG CRAMPS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
LEG PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
LEG PAIN (RELATED TO HERNIATED DISC) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
LICHEN PLANUS MOUTH + TONGUE (Gastrointestinal disorders) | 0 (0) | 1 (1)
LLQ ABDOMINAL PAIN WITH BM (Gastrointestinal disorders) | 0 (0) | 1 (1)
LOOSE STOOL (Gastrointestinal disorders) | 1 (1) | 2 (3)
LOW BLOOD COUNT (Investigations) | 1 (1) | 0 (0)
LOW BONE DENSITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LOWBACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LOWER BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
LOWER LEG SWELLINGW (Vascular disorders) | 0 (0) | 1 (1)
LOWERBACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
LOWGRADE FEVER (General disorders) | 0 (0) | 1 (1)
LYMPHADENITIS RIGT NECK (Vascular disorders) | 1 (1) | 0 (0)
MASS FOUND ON CRX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MORE FREQUENT HEADACHES (Nervous system disorders) | 0 (0) | 1 (1)
MUCUS/COUGHING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
MULTIPLE POLYPS (<4MM) IN FLEX SIGMOIDOSCOPY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MULTIPLE POLYPS IN THE COLONOSCOPY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MUSCLE SPASMS IN BACK (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL ACHE ARM LEFT (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL ACHINESS, TIGHTNESS - KNEES (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL ANKLE INJURY, LEFT, R/T MISSTEP (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL BACK SPASM (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL BACK STRAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL BILATERAL LOWER EXTREMITY FATIGUE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL BILATERAL THIGH CRAMPS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL BUMP INTERIOR TO LEFT ELBOW (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL CRAMPS THIGH RIGHT (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL CRAMPS THIGHS BILATERAL (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL FOOT PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL GANGLION CYST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MUSCULOSKELETAL INCREASED BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL L2, L3 DISKS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL LEFT HIP PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL LEFT INGUINAL HERNIA, RECURRENT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL MIDDLE FINGER CYST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MUSCULOSKELETAL MINOR BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL MUSCLE PAIN, RIGHT LEG (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL MUSCLE SORENESS - R FOREMARM (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL MUSCLE WEAKNESS/SORENESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL NECK PAIN FROM FALL (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL OLECRANON BURSITIS/CELLULITIS/ELBOW SWELLING (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN - BILATERAL KNEE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL PAIN - RIGHT KNEE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL RIGHT KNEE SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL RIGHT KNEE TORN MENISCUS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL RIGHT ROTATOR CUFF, PAIN JOINT FUNCTION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL SCIATICA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL SHOULDER PAIN CONTINUES (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL SPRAINED ANKLE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL TAILBONE INJURY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL THIGH CRAMPS BILATERAL (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL TORN ROTATOR CUFF, LEFT (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL UNSTEADY GAIT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL VENTRAL HERNIA X 2 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 16 (18) | 11 (16)
NAUSEA 5 EPISODES (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA AFTER COLONOSCOPY (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA AND BELCHING (Gastrointestinal disorders) | 1 (2) | 0 (0)
NAUSEA NAUSEA/DIARRHEA/HEADACHE (Gastrointestinal disorders) | 1 (3) | 0 (0)
NAUSEA POST SURGICAL (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA RELATED TO NEW MEDICINE GLUCOPHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
NECK AND SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
NECK PAIN, INJURY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
NEUROLOGY - DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0)
NEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1)
NEUROPATHY/SENSORY; TINGLING IN FINGERS (Nervous system disorders) | 1 (1) | 0 (0)
NOSEBLEED (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
NUMBNESS/TINGLING OF RIGHT ARM (Nervous system disorders) | 1 (1) | 0 (0)
OA PAIN (HIPS) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OCC. CHEST TIGHTNESS (Cardiac disorders) | 0 (0) | 1 (1)
OCCULAR MIGRAIN (Nervous system disorders) | 1 (1) | 0 (0)
OLECRANON BURSITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ORAL HAD BUMP ON SURFACE OF TONGUE (Gastrointestinal disorders) | 1 (1) | 0 (0)
ORAL SORE NEAR RIGHT INCISOR (Gastrointestinal disorders) | 1 (1) | 0 (0)
ORAL SORENESS, UPPER RIGHT GUM WHERE PREVIOUSLY BAD TOOTH REMOVED (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL SORES (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL* BLISTER ROOF OF MOUTH (Gastrointestinal disorders) | 1 (1) | 0 (0)
ORAL* CANKER SORES (Gastrointestinal disorders) | 1 (1) | 0 (0)
ORAL* CANKER SORES ON TONGUE (Gastrointestinal disorders) | 1 (1) | 0 (0)
ORAL* CHAPPED LIPS (Gastrointestinal disorders) | 1 (2) | 0 (0)
ORAL* COLD SORES, LIPS (Gastrointestinal disorders) | 3 (3) | 0 (0)
ORAL* CONT. ESOPHAGEAL IRRITATION/SORE THROAT WITH DIFFICULTY SWALLOWING POSSIBLY DUE TO ROSACEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ORAL* DIFFICULTY SWALLOWING POSSIBLY DUE TO ROSACEA MEDS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL* DISCOLORING OF TEETH (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL* DISCOMFORT MOUTH, POST DENTAL WORK (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL* DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 1 (1)
ORAL* DRY THROAT (Gastrointestinal disorders) | 1 (1) | 0 (0)
ORAL* DRY THROAT/MOUTH (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL* DYSGEUSIA/TASTE DISTURBANCE (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL* DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL* EXACERBATION/ LICHEN PLANUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ORAL* GINGIVITIS FROM TEETH SCALING (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL* GUM PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
ORAL* HYPERTROPHY, LUMP LEFT UPPER GUM (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL* INCREASED SALIVA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ORAL* INTERMITTENT ORAL ULCERS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL* LESION (Gastrointestinal disorders) | 1 (1) | 0 (0)
ORAL* LESION ON LOWER LIP (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL* MOUTH DRYNESS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL* MOUTH SORE (Gastrointestinal disorders) | 1 (1) | 0 (0)
ORAL* MOUTH SORES (Gastrointestinal disorders) | 1 (1) | 0 (0)
ORAL* PAIN - SOFT PALATE POST SURGICAL (Gastrointestinal disorders) | 1 (1) | 0 (0)
ORAL* PAIN IN MOUTH POST PERIODONTAL SURGERY (Gastrointestinal disorders) | 1 (1) | 0 (0)
ORAL* PAIN RIGHT UPPER MOLAR (Gastrointestinal disorders) | 1 (1) | 0 (0)
ORAL* PRE-ABSCESS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ORAL* SORE GUM - RIGHT (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL* SORE THROAT (Gastrointestinal disorders) | 0 (0) | 4 (5)
ORAL* SORENESS (Gastrointestinal disorders) | 1 (1) | 1 (1)
ORAL* THROAT DRYNESS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL* THROAT IRRITATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL* TOOTH PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
ORAL* ULCERS (Gastrointestinal disorders) | 1 (2) | 0 (0)
ORAL* YEAST INFECTION (Infections and infestations) | 1 (1) | 0 (0)
OTHER CONJUNCTIVITIS, WITH OP EYE SURGERY (Eye disorders) | 1 (1) | 0 (0)
OTHER* + + PITTING BILATERAL ANKLE EDEMA (General disorders) | 1 (1) | 0 (0)
OTHER* 1 CM LESION ON RT. HAND (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER* 2 LUMPS IN GROIN AREA (SIZE 2 X 2 CM) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER* ABCESS OF FINGER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER* ABDOMINAL BLOATING (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER* ACTINIC KERATOSIS REMOVED (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER* ADENOMA POLYP (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER* ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER* ALLERGIES (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 2 (2)
OTHER* ALLERGY PET (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER* ALLERGY SYMPTOMS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (5)
OTHER* ALTERED TASTE (Nervous system disorders) | 0 (0) | 1 (1)
OTHER* ALTERED TASTE CHOCOLATE (Nervous system disorders) | 0 (0) | 1 (1)
OTHER* ANAL FISTULA (Gastrointestinal disorders) | 1 (2) | 0 (0)
OTHER* ANAL FISTULA, SURG REPAIR (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER* ARTHRALGIA LEFT ANKLE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER* ARTHRALGIA LEFT ELBOW (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER* ARTHRALGIA LEFT SHOULDER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER* ARTHRALGIA LEFT WRIST (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER* ARTHRALGIA LOWER BACK (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER* ARTHRALGIA NECK (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER* BACK PAIN AND DIARRHEA (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
OTHER* BACK STRAIN (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
OTHER* BAD COLD X 3 WKS (General disorders) | 1 (1) | 0 (0)
OTHER* BASAL CELL CARCINOMA LEFT CLAVICLE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER* BASAL CELL CARCINOMA LEFT JAW (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER* BILATERAL FOOT EDEMA R>L (General disorders) | 0 (0) | 1 (1)
OTHER* BILATERAL FOOT TINGLING (Nervous system disorders) | 0 (0) | 1 (1)
OTHER* BILATERAL LOWER EXTREMEITY EDEMA (General disorders) | 0 (0) | 1 (1)
OTHER* BIOPSY OF SKIN NEOPLASM, ABD. CYST AND THIGH (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER* BLADDER POLYP (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER* BLEPHARITIS (Eye disorders) | 0 (0) | 1 (1)
OTHER* BLOATING (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER* BLOATING, HX IBS (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER* BLOODY MUCOUS/ EXPECTORATED (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER* BODY ACHES (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
OTHER* BODY ACHES GENERAL (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
OTHER* BODY ODOR DIFFERENT (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER* BOIL ON COCCYX (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER* BONE SPUR/HEEL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER* BRACHY THERAPY FOR PROSTATE CA (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER* BREAST BIOPSY (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER* BREAST LUMP (FNA NEG) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER* BROKEN RIGHT UPPER ARM AND RIGHT FOOT R/T FALL (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER* BURSITIS - SHOULDER (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
OTHER* BURSITIS IN RIGHT SHOULDER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER* BURSITIS RIGHT SHOULDER (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
OTHER* BURSITIS-ELBOW (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER* CARPAL TUNNEL SYNDROME BILATERAL (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER* CELLULITIS RIGHT KNEE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER* CHEST X-RAY ABNORMAL, RIGHT UPPER LOBE LESION (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER* CHILLS, JOINT PAIN, SKIN IS SENSITIVE (General disorders) | 0 (0) | 1 (3)
OTHER* CLAUDICATION (Cardiac disorders) | 1 (1) | 0 (0)
OTHER* COCCYX INJURY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER* COLD SORE (NOSE) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER* CONJUNCTIVITIS (ALLERGIC) (Eye disorders) | 0 (0) | 1 (1)
OTHER* COPD EXACERBATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
OTHER* CRAMPING (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER* CUTS TAKE LONGER TO HEAL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER* CYST IN GROIN WITH INFECTION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER* CYST ON BACK, DRAINED 10/10/00 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER* DECREASED LIBIDO (Psychiatric disorders) | 1 (1) | 1 (1)
OTHER* DECREASED THYROID FUNCTION, THIN HAIR, DECREASED TEMP, DRY SKIN (Endocrine disorders) | 1 (1) | 0 (0)
OTHER* DEGENERATIVE JOINT DISEASE-RIGHT GREAT TOE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER* DEGENERATIVE JOINT DISEASE; LOW BACK (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER* DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER* DEPRESSION (Psychiatric disorders) | 1 (1) | 2 (2)
OTHER* DEPRESSION - RECURRANCE (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER* DEPRESSIVE SX, RELATIONSHIP CONCERNS (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER* DIABETES (Endocrine disorders) | 2 (2) | 0 (0)
OTHER* DIABETIC NEUROPATHY (Endocrine disorders) | 0 (0) | 1 (1)
OTHER* DIFFICULTY SWALLOWING(DYSPHAGIA) (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER* DISCOMFORT - RIGHT LEG (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER* DISCOMFORT LEFT EAR (Ear and labyrinth disorders) | 0 (0) | 1 (1)
OTHER* DISCOMFORT LEFT KNEE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER* DISCOMFORT POST PROSTATE BIOPSY (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER* DRY EYES (Eye disorders) | 1 (1) | 0 (0)
OTHER* DX METRORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER* DX OF DIABETES (Endocrine disorders) | 1 (1) | 0 (0)
OTHER* DYSGEUSIA (Nervous system disorders) | 0 (0) | 1 (1)
OTHER* DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER* DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER* DYSPLASIA PROSTATE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER* EAR DISCHARGE (Ear and labyrinth disorders) | 0 (0) | 1 (1)
OTHER* EAR PAIN AND PRESSURE (Ear and labyrinth disorders) | 1 (1) | 0 (0)
OTHER* EDEMA (General disorders) | 1 (1) | 0 (0)
OTHER* EDEMA LEFT EXTREMITY (General disorders) | 1 (1) | 0 (0)
OTHER* ELEVATED BLOOD PRESSURE/ SINGLE EVENT 9/00 (Cardiac disorders) | 0 (0) | 1 (1)
OTHER* ELEVATED BLOOD PRESSURE; SINGLE 9/00 (Cardiac disorders) | 0 (0) | 1 (1)
OTHER* EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER* ENDOCRINE -- HOT FLASHES (Endocrine disorders) | 1 (1) | 0 (0)
OTHER* ENLARGED PROSTATE, PT PLACED ON PROZOSIN (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER* EPISCLERITIS (Eye disorders) | 0 (0) | 1 (1)
OTHER* ERECTILE DYSFUNCTION, INCREASED SEVERITY OVER TIME (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER* ERODED ESOPHAGUS/GERD (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER* ESOPHAGEAL SPASM (Gastrointestinal disorders) | 1 (2) | 1 (1)
OTHER* ESOPHAGEAL STRICTURE (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER* ESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER* F/U 6MO CT (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER* FEELS "FUZZY" IN HER HEAD (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER* FLOATER D/T DIABETIC RETINOPATHY (Eye disorders) | 0 (0) | 1 (1)
OTHER* FOOD POISONING (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER* FOOD POISONING: DIARRHEA. VOMITTING (Gastrointestinal disorders) | 1 (2) | 0 (0)
OTHER* FORGETFULNESS, LOSS OF TRAIN OF THOUGHT (Nervous system disorders) | 0 (0) | 1 (1)
OTHER* GALLSTONES (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER* GASTRITIS, DEHYDRATION, RESPIRATORY TRACT INFECTION, FATIGUE (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER* GENERAL ACHES (General disorders) | 1 (1) | 0 (0)
OTHER* GENERAL BODY ACHES (General disorders) | 0 (0) | 1 (1)
OTHER* GENITOURINARY "TWINGE" RIGHT TESTICLE (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER* GENITOURINARY BLADDER SPASMS (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER* GENITOURINARY, LEFT TESTICLE TENDER/SWOLLEN (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER* GENITOURINARY/ VAGINITIS (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER* GERD (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER* GLAUCOMA (Eye disorders) | 1 (1) | 0 (0)
OTHER* GLAUCOMA INCREASED (Eye disorders) | 1 (1) | 0 (0)
OTHER* GRIEF/DEPRESSION FM. DEATH (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER* GU - URINARY FREQUENCY (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER* GU BLADDER SPASMS (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER* HARDER STOOLS (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER* HEAD GETS COLD (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER* HEARTBURN (Gastrointestinal disorders) | 7 (15) | 7 (9)
OTHER* HEARTBURN 2X WEEKLY (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER* HEARTBURN 3 TIMES A WEEK (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER* HEARTBURN X 3 EPISODES (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER* HEARTBURN X5 EPISODES (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER* HEARTBURN, 3-4 EPISODES/WEEK (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER* HEARTBURN, INCREASE? (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER* HEME + X3 (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER* HEMOPTISIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER* HOT AND SWEATY (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER* HOT FLASHES, STOPPED HRT MEDS (Vascular disorders) | 0 (0) | 1 (1)
OTHER* HSV OUTBREAK (Infections and infestations) | 1 (2) | 0 (0)
OTHER* HT OF GASTRIC ULCERS (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER* HTN (Cardiac disorders) | 1 (1) | 0 (0)
OTHER* HTN (R/T STRESS AND WEIGHT) (Cardiac disorders) | 0 (0) | 1 (1)
OTHER* IGA GLOMERULONEPHRITIS (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER* IMPOTENCE (Reproductive system and breast disorders) | 1 (1) | 1 (1)
OTHER* INCONTINENCE (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER* INCREASE IN DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER* INCREASE IN TREMORS (Nervous system disorders) | 0 (0) | 1 (1)
OTHER* INCREASED DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER* INCREASED GAS WITH EATING (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER* INCREASED PSA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER* INCREASED STRESS (General disorders) | 1 (1) | 2 (2)
OTHER* INCREASED URINARY URGENCY (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER* INCREASING INCONTINENCE (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER* INFECTION SINUS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER* INSOMNIA (Psychiatric disorders) | 3 (7) | 0 (0)
OTHER* INSOMNIA - TROUBLE SLEEPING (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER* INSOMNIA INCREASE (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER* IRRITABILITY (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER* IRRITATED THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER* ITCHY EYES (Eye disorders) | 0 (0) | 1 (1)
OTHER* KIDNEY STONES (Renal and urinary disorders) | 1 (2) | 0 (0)
OTHER* KNEE STRAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER* LACERATION, ER VISIT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER* LAPSES IN CONCENTRATION (Nervous system disorders) | 0 (0) | 1 (1)
OTHER* LEFT ARM FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER* LEFT BREAST NODULE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER* LEFT FOOT ARCH BRUISE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER* LEFT NIPPLE IRRITATED (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER* LESION ON RIGHT THIGH (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER* LETHARGY (General disorders) | 0 (0) | 1 (1)
OTHER* LIGHTHEADEDNESS (Nervous system disorders) | 0 (0) | 1 (2)
OTHER* LOOSE SPHINCTER RECTURM-SEEPAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER* LOOSE STOOL (Gastrointestinal disorders) | 1 (1) | 1 (1)
OTHER* LOWER EXTREMITY EDEMA (General disorders) | 1 (1) | 0 (0)
OTHER* LOWER EXTREMITY EDEMA - BILATERAL (General disorders) | 0 (0) | 1 (1)
OTHER* LUMP IN RIGHT GROIN, LYMPHADENOPATHY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER* LUNG CANCER LEFT HILAR MASS SQUAMOUS CELL LYMPH NODE THORAX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER* MECHANICAL FALL WITH LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER* MENOPAUSE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER* MILD PARESTHESIA (Nervous system disorders) | 1 (1) | 0 (0)
OTHER* MILD PARESTHESIA, BILATERAL ARMS (Nervous system disorders) | 0 (0) | 1 (1)
OTHER* MODERATE PARESTHESIA (Nervous system disorders) | 1 (1) | 0 (0)
OTHER* MODERATE PARESTHESIA IN RIGHT HAND (Nervous system disorders) | 1 (1) | 0 (0)
OTHER* MOUTH COLD SORE (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER* MUCLE PULLED BACK (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER* NAIL AVULSION, LEFT HALLUX NAIL (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER* NASAL DISCHARGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER* NERVOUS REACTION (Nervous system disorders) | 0 (0) | 1 (1)
OTHER* NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER* NUMBNESS LEFT PINNA (Nervous system disorders) | 0 (0) | 1 (1)
OTHER* OCCASIONAL BRUISING (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER* OCCASIONAL LOSS OF ERECTION DURING INTERCOURSE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER* OCULAR - DRY MACULAR DEGENERATION (Eye disorders) | 0 (0) | 1 (1)
OTHER* OCULAR - INCREASE INTRAOCULAR PRESSURE LEFT EYE (Eye disorders) | 1 (1) | 0 (0)
OTHER* OCULAR/VISUAL MYOPIA (Eye disorders) | 1 (1) | 0 (0)
OTHER* ORAL SORENESS; ABCESS LOWER GUM (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER* OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER* OSTEOPOROSIS-LEFT WRIST (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER* PAIN-LEFT ANKLE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER* PARESTHESIA (Nervous system disorders) | 0 (0) | 1 (1)
OTHER* PARESTHESIA GREAT TOE RIGHT (Nervous system disorders) | 0 (0) | 1 (1)
OTHER* PARESTHESIA TOES (Nervous system disorders) | 0 (0) | 1 (1)
OTHER* PARESTHESIA TOES LEFT FOOT (Nervous system disorders) | 0 (0) | 1 (1)
OTHER* PARESTHESIA-LEFT ARM (Nervous system disorders) | 1 (1) | 0 (0)
OTHER* PERIANAL ABSCESS (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER* PERIANAL SWELLING (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER* PHLEBITIS LEFT FOREARM (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER* PHLEBITIS SUPERFICIAL LEFT FOREARM (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER* PLANTAR FASCIITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER* PLANTAR FASCIITIS LEFT FOOT (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER* POST NASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER* PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
OTHER* PROSTATIC ADENOCARCINOMA DX 7/01/03 BY BX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER* PRURITIUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER* PRURITIUS LEGS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER* PRURITIUS, HIPS AND BELLY (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER* PRURITUS, INTERMITTENT, BELLY, HIPS, LEGS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER* PRURITUS, INTERMITTENT, HIPS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER* RECTAL BOIL (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER* RECTAL MOISTNESS (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER* RECTAL URGENCY (Gastrointestinal disorders) | 0 (0) | 1 (2)
OTHER* RECTOCELE, VAGINAL (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER* RED LINE ON TOE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER* REDDENED EYES (Eye disorders) | 1 (1) | 0 (0)
OTHER* REMOVAL OF SHRAPNEL (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER* RETINA EDEMA, POST OP (Eye disorders) | 1 (1) | 0 (0)
OTHER* RETINAL TEAR LEFT EYE (Eye disorders) | 0 (0) | 1 (2)
OTHER* RIGHT EAR PRESSURE (Ear and labyrinth disorders) | 1 (1) | 0 (0)
OTHER* RIGHT EYE BLURRINESS (Eye disorders) | 0 (0) | 1 (1)
OTHER* RIGHT GREAT TOE WITH REDDISH SPOT (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER* RIGHT INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER* ROOT CANAL X3 (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER* RUNNY NOSE (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
OTHER* SCRATCHY THROAT/SNIFFLES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER* SHADOW IN LEFT LUNG, POSS. BENIGN TUMOR OR SCAR TISSUE. CT 3/10/04 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER* SINUS INFECTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER* SINUS PROBLEM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER* SKIN LESION LEFT FOREARM (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER* SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER* SLEEPY (General disorders) | 0 (0) | 1 (1)
OTHER* SMALL GOITER (Endocrine disorders) | 0 (0) | 1 (1)
OTHER* SNIFFLES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER* SOB CHEST TIGHTNESS, POSSIBLE GERD SX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER* SORE SHOULDER RELATED TO PAST BREAK (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER* SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
OTHER* SPIDER BITE (LEG) SWELLING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER* STIFF FINGERS RIGHT. GOLF? (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER* STOMACH CRAMPING (Gastrointestinal disorders) | 0 (0) | 1 (2)
OTHER* STRAIN LEFT ARM (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER* STRESS, INCREASED (General disorders) | 0 (0) | 1 (1)
OTHER* SUBORBITAL EDEMA, RIGHT EYE (Eye disorders) | 0 (0) | 1 (1)
OTHER* SYNCOPE X 1 (Nervous system disorders) | 0 (0) | 1 (1)
OTHER* TEARY/WATERY EYES (Eye disorders) | 0 (0) | 1 (1)
OTHER* TENDON, BRUISED RIGHT ELBOW (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER* THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER* TINGLING LEFT FOOT (Nervous system disorders) | 1 (1) | 0 (0)
OTHER* TINGLING TONGUE (Nervous system disorders) | 0 (0) | 1 (1)
OTHER* TURP (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER* ULCERATION, RT LOWER EXTREMITY (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER* UNSTEADY GAIT (Nervous system disorders) | 0 (0) | 1 (1)
OTHER* URGENCY TO URINATE WITH BURNING AT TIMES (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER* URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER* URINARY URGENCY (Renal and urinary disorders) | 1 (1) | 1 (1)
OTHER* URINATION PAIN (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER* URTICARIA (Immune system disorders) | 0 (0) | 1 (1)
OTHER* UTERINE POLYP (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER* VAGINAL ITCHING (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER* VERY LOOSE STOOL (Gastrointestinal disorders) | 0 (0) | 1 (4)
OTHER* VOICE CHANGE - HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER* WHITE BLOOD CELL COUNT INCREASE (Investigations) | 1 (1) | 0 (0)
OTOTOXICITY* LEFT EAR (Ear and labyrinth disorders) | 1 (1) | 0 (0)
OTOTOXICITY* R/EAR CLOGGED (Ear and labyrinth disorders) | 1 (1) | 0 (0)
OTOTOXICITY* TINNITUS LEFT EAR (Ear and labyrinth disorders) | 1 (1) | 0 (0)
PAIN (General disorders) | 1 (1) | 0 (0)
PAIN AND LOCAL SWELLING, UPPER LEFT MOLAR (Gastrointestinal disorders) | 1 (1) | 0 (0)
PAIN FROM KIDNEY STONES (Renal and urinary disorders) | 0 (0) | 1 (1)
PAIN IN LOWER CALF (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* "VAGUE PAIN" WEAKNESS LEFT LEG (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
PAIN* ALL OVER BODY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* ANKLE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* ARTHRALAGIA LEFT HAND (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* BACK (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (7)
PAIN* BACK INCREASING (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* BACK INTERMITTENT (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* BACK LOWER LEFT (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
PAIN* BACK PAIN WHILE EXERCISING (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* BACK X2 EPISODES (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* BACK, MUSCLE SPASM (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* BILATERAL KNEE SORENESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* BILATERAL SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* BODY ACHES (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* BREAST TENDERNESS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
PAIN* CERVICAL - NECK (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* CHEST (Cardiac disorders) | 2 (2) | 0 (0)
PAIN* CHEST DISCOMFORT (Cardiac disorders) | 0 (0) | 1 (1)
PAIN* CHEST; EXACERBATION OF PREVIOUS CONDITION (Cardiac disorders) | 1 (1) | 0 (0)
PAIN* EAR (Ear and labyrinth disorders) | 0 (0) | 1 (1)
PAIN* EAR ACHE (Ear and labyrinth disorders) | 1 (1) | 1 (1)
PAIN* EAR PAIN (Ear and labyrinth disorders) | 1 (1) | 0 (0)
PAIN* FINGER PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* FLANK PAIN, KIDNEY STONES (Renal and urinary disorders) | 1 (1) | 0 (0)
PAIN* FOOT PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* FOOT PAIN/SORE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* FROM SEED IMPLANT FOR PROSTATE CA (Surgical and medical procedures) | 1 (1) | 0 (0)
PAIN* GAS (Gastrointestinal disorders) | 1 (2) | 0 (0)
PAIN* GENERAL MUSCLE/JOINT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* GREAT TOE RIGHT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* GREAT TOES PAINFUL (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* GROIN PAIN/ PUBIC BONE WITH LONG SITTING (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* HANDS JOINT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
PAIN* HEADACHE SINUS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* HIPS/BACK (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* IN CHEST R/T FALL (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* IN FRONT OF LEFT UPPER THIGH (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* JOINTS INCREASING (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* JOINTS OF LEFT SIDE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* KNEE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* KNEE LIGAMENT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* KNEE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* LEFT ACHILLES (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* LEFT ANKLE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* LEFT ARM (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* LEFT ARM W/TINGLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* LEFT FOOT (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* LEFT HAND (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* LEFT HEEL (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* LEFT HEEL BONE SPUR (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* LEFT HIP (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
PAIN* LEFT KNEE (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
PAIN* LEFT LOWER EXTREMITY CLAUDICATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* LEFT NECK (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* LEFT SHOULDER (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
PAIN* LEFT TESTICLE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PAIN* LEFT THUMB (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* LEG CRAMPS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
PAIN* LOW BACK (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (5)
PAIN* LOWER BACK STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* MILD BACK PAIN "BURNING" (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* MUSCLE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* MUSCLE ACHES (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* MUSCLE STRAIN (PAIN) IN LOWER BACK (OCCASIONAL) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* MUSCLE STRAIN/SPASM (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
PAIN* MVA - CHEST WALL PN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* MVA BACK PN/LEG PN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* NECK (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
PAIN* NECK & BACK (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* NECK & UPPER CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
PAIN* NECK, INJURY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* PAIN IN LEFT LEG AND KNEE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* PELVIC CRAMPING (Gastrointestinal disorders) | 0 (0) | 1 (8)
PAIN* POST - SURGICAL (Surgical and medical procedures) | 1 (1) | 0 (0)
PAIN* POST HERNIA REPAIR (Surgical and medical procedures) | 0 (0) | 1 (1)
PAIN* POST ORAL SURGERY (Surgical and medical procedures) | 1 (1) | 0 (0)
PAIN* POST ROOT CANAL (Surgical and medical procedures) | 2 (3) | 0 (0)
PAIN* POST SURGICAL (Surgical and medical procedures) | 1 (1) | 0 (0)
PAIN* POST TOOTH EXTRACTION (Surgical and medical procedures) | 2 (2) | 0 (0)
PAIN* PULLED MUSCLE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* RECTAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
PAIN* RIGHT BACK PAIN, INJURY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* RIGHT BREAST (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PAIN* RIGHT BUTTOCKS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* RIGHT FLANK (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* RIGHT GREAT TOE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* RIGHT HEEL (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
PAIN* RIGHT HEEL - PLANTAR FASCIITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* RIGHT HIP AND KNEE (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
PAIN* RIGHT KNEE (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
PAIN* RIGHT KNEE - INCREASE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* RIGHT LEG PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* RIGHT LOWER BACK (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* RIGHT LOWER BACK AND LEFT KNEE PAIN (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
PAIN* RIGHT LOWER BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* RIGHT SHOULDER (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
PAIN* RIGHT SHOULDER BLADE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* RIGHT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* RIGHT SIDED PAIN AFTER EXERCISE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* RLQ (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* RT LEG SECONDARY TO FALL (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* RT. RING FINGER, RT PINKY NUMBNESS/TINGLING (Nervous system disorders) | 0 (0) | 1 (1)
PAIN* RUQ PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
PAIN* SCIATICA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* SCORPION BITE RIGHT FOREARM (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PAIN* SHIN LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PAIN* SHOULDERS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
PAIN* SORE KNEE (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
PAIN* SORE LEFT BIG TOE - GOUT? (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
PAIN* SORE LEFT SHOULDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* SORE ON THUMB (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* SORE RT. KNEE, INCREASED PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
PAIN* SPRAINED ANKLE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN* STERNAL PAIN/BURNING SENSATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PAIN* STIFF NECK R/T HEAD BUMP IN BATH (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* STIFFNESS & PAIN IN WRIST (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
PAIN* STOMACH (Gastrointestinal disorders) | 0 (0) | 1 (2)
PAIN* TAILBONE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN* TESTICLE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PAIN* TESTICULAR SORENESS & SWELLING (Reproductive system and breast disorders) | 1 (2) | 0 (0)
PAIN* TOOTH (Gastrointestinal disorders) | 1 (1) | 0 (0)
PAIN* UPPER RIGHT QUADRANT (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN/MUSCULOSKELETAL/SOFT TISSUE; EXTREMITY - UPPER LEFT SHOULDER ROTATOR CUFF TEAR REAPAIR (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PARKINSONS DISEASE (Nervous system disorders) | 0 (0) | 1 (1)
PERIPHERAL NERVOUS SYSTEM* (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL NERVOUS SYSTEM* ARMS TINGLE/GO NUMB (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL NERVOUS SYSTEM* HAND TREMBLINGS (Nervous system disorders) | 0 (0) | 1 (1)
PERIPHERAL NERVOUS SYSTEM* HAND TREMOR (Nervous system disorders) | 0 (0) | 1 (1)
PERIPHERAL NERVOUS SYSTEM* MILD PARESTHESIA (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL NERVOUS SYSTEM* MILD PARESTHESIA BOTH HANDS (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL NERVOUS SYSTEM* NEURO SCIATIC RIGHT LEG (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL NERVOUS SYSTEM* NEURO SCIATICA RIGHT LEG (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL NERVOUS SYSTEM* OLD INJURY (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL NERVOUS SYSTEM* PARESTHESIA (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL NERVOUS SYSTEM* PARESTHESIA BILAT TINGLING IN SHOULDERS (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL NERVOUS SYSTEM* PARESTHESIA L/HAND NUMBNESS (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL NERVOUS SYSTEM* PARESTHESIA LEFT SHOULDER PINCHED NERVE (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL NERVOUS SYSTEM* PERESTHESIA, FEET, INCREASED FROM BASELINE (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL NERVOUS SYSTEM* RIGHT FOOT TOE NUMBNESS (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL NERVOUS SYSTEM* RIGHT LEG NUMBNESS (Nervous system disorders) | 0 (0) | 1 (1)
PERIPHERAL NERVOUS SYSTEM* SLIGHT TINGLING/NUMBNESS HANDS/WRIST (Nervous system disorders) | 0 (0) | 1 (1)
PERIPHERAL NERVOUS SYSTEM* SPINAL STENOSIS (Nervous system disorders) | 1 (1) | 0 (0)
POSSIBLE FUNGAL INFECTION (SCALP) (Infections and infestations) | 0 (0) | 1 (1)
POSSIBLE RENAL CALCULUS (TOOK 1 VICODINE) (Renal and urinary disorders) | 1 (1) | 0 (0)
POST NASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PROCTALGIA FUGAX (Gastrointestinal disorders) | 0 (0) | 1 (1)
PROTRUDING AND TENDER HEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 0 (0)
PSEDOTUMOR EYE WILL F/U IN 6 MONTHS (Eye disorders) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
RASH ABDOMINAL (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH BODY AND EXTREMITIES (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH BUMPS ON SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH EXACERBATION OF SEASONAL ITCHY RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH FACE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH HANDS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH ITCH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH RIGHT CHEEK (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH RIGHT FOOTECZEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH RIGHT FOREARM (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH RIGHT LEG (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH SHINGLES (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
RASH SKIN RIGHT UPPER ARM (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RASH URTICARIA RIGHT BUTTOCK (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
REFLUX (Gastrointestinal disorders) | 2 (2) | 3 (4)
REFLUX ACID (Gastrointestinal disorders) | 1 (1) | 0 (0)
REFLUX ACID REFLUX (Gastrointestinal disorders) | 0 (0) | 2 (2)
REFLUX ACID REFLUX 2-3 EPISODES/WK (Gastrointestinal disorders) | 0 (0) | 1 (1)
REFLUX ACID REFLUX DAILY (Gastrointestinal disorders) | 0 (0) | 1 (1)
REFLUX GASTRIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
REFLUX GERD (Gastrointestinal disorders) | 1 (1) | 0 (0)
REFLUX GERD EPISODE (Gastrointestinal disorders) | 1 (2) | 0 (0)
REFLUX GERD EPISODIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
REFLUX GERD, INCREASED SEVERITY OF EPISODES (Gastrointestinal disorders) | 0 (0) | 1 (1)
REFLUX INCREASED GERD, NUMBER OF EPISODES (Gastrointestinal disorders) | 1 (1) | 0 (0)
RELEASE OF CARPAL TUNNEL IN RIGHT HAND (Surgical and medical procedures) | 1 (1) | 0 (0)
REMOVAL OF PINS FROM PRIOR BUNIONECTOMY RIGHT FOOT (Surgical and medical procedures) | 0 (0) | 1 (1)
REMOVAL PRE-CAN SK. (Surgical and medical procedures) | 1 (2) | 0 (0)
RESPIRATORY ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY ALLERGIES/ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY ASTHMA FLARE UP (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
RESPIRATORY ASTHMA FLARE-UP, WHEEZING, SOB (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY BRONCHIAL ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
RESPIRATORY CHEST COLD SX, DX WITH PNEUMONIA RIGHT LUNG (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY CHEST CRX, PNEUMONIA RIGHT LUNG (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY CHOKING ON SALIVA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY CHRONIC RHINITIS CONTINUES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY COLD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY COLD SYMPTOMS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY COLD SYMPTOMS: NASAL DRAINAGE, CONGESTION, COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY COPD EXACERBATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
RESPIRATORY DIAPHRAGM DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY DX WITH BRONCHIAL PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY DYSPNEA ON EXERTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY INFECTION, BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY RHINITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY SHORT OF BREATH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
RESPIRATORY SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
RESPIRATORY SHORTNESS OF BREATH 2X (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY SINUS INFECTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
RESPIRATORY SOB 6 EPISODES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY SOB WITH EXERTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY SOB WITH HEAVY EXERCISE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY STUFFY NOSE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY UPPER RESPIRATORY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY UPPER, INFLUENZA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY UPPER, SINUS PROBLEM ALLERGY RELATED (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY URI (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RIGHT ANKLE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
RIGHT EAR SENSORAL HEARING LOSS -- AGE RELATED PER ENT MD (Ear and labyrinth disorders) | 0 (0) | 1 (1)
RIGHT ELBOW TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
RIGHT RENAL CYST (Gastrointestinal disorders) | 0 (0) | 1 (1)
RIGHT SIDE ABOVE EAR (Ear and labyrinth disorders) | 1 (1) | 0 (0)
RIGHT TELBOW TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
RINORRHEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ROSACASE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RT ELBOW FX (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SEASONAL ALLERGIES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
SERUM GLUCOSE (Investigations) | 1 (1) | 0 (0)
SEVERE BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SEXUAL DYSFUNCTION (Reproductive system and breast disorders) | 0 (0) | 1 (1)
SHINGLES (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SHOULDER PAIN OLD INJURY FLAIR UP (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SIGNIFICANT OTHER PERCEPTION OF CHANGE IN HEARING (Ear and labyrinth disorders) | 0 (0) | 1 (1)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 2 (2)
SINUS CONGESTION & ALLERGIES (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SINUS CONGESTION ALLERGIES (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
SINUS CONGESTION CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SINUS CONGESTION HEAD CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SINUS CONGESTION SINUS INFECTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SINUS CONGESTION SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SINUS DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
SINUS HEADACHE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SINUS INFECTION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
SKIN LESION REMOVED (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKIN RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SLEEP APNEA (Nervous system disorders) | 1 (1) | 0 (0)
SLIGHT QUEEZY STOMACH (Gastrointestinal disorders) | 1 (1) | 0 (0)
SMALL OUTBREAKS OF PUSTULES UNDER NOSTRILS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SORE THROAT, COUGH, BODY ACHES, 103 TEMP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SORE THROAT, MUCUS/COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SPINNING (Nervous system disorders) | 1 (1) | 0 (0)
SPRAINED ANKLE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SQUAMOUS CELL REMOVAL (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
STOMACH ACHE (Gastrointestinal disorders) | 0 (0) | 1 (1)
STOMACH FLU (Gastrointestinal disorders) | 1 (1) | 0 (0)
STOMACH PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
STOMACH UPSET AND HEARTBURN (Gastrointestinal disorders) | 1 (2) | 0 (0)
STOMACH VIRUS (VIRAL GASTROECTERITIS) (Gastrointestinal disorders) | 1 (1) | 0 (0)
STOOL* BLACK (Gastrointestinal disorders) | 0 (0) | 1 (1)
STOOL* CLEAR RECTAL DISCHARGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
STOOL* DISCOLORED (Gastrointestinal disorders) | 0 (0) | 1 (1)
STOOL* HARD (Gastrointestinal disorders) | 0 (0) | 1 (1)
STOOL* HIGHER FREQUENCY (Gastrointestinal disorders) | 1 (1) | 0 (0)
STOOL* LOOSE (Gastrointestinal disorders) | 2 (2) | 1 (1)
STOOL* LOOSE, 2-3 DAYS/WEEK (Gastrointestinal disorders) | 1 (1) | 0 (0)
STOOL* LOOSER (Gastrointestinal disorders) | 1 (1) | 0 (0)
STOOL* SOFT WITH ABDOMINAL CRAMPS (Gastrointestinal disorders) | 1 (1) | 0 (0)
STOOL* TARRY (Gastrointestinal disorders) | 1 (1) | 0 (0)
STREP THROAT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SUBCONJUNCTIVAL HEMORRHAGE (Eye disorders) | 1 (1) | 0 (0)
SURGERY* CABG WOUNDS (CORONARY ARTERY BYPASS GRAFT) (Surgical and medical procedures) | 1 (1) | 0 (0)
SURGERY* CHOLESYSTECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
SURGERY* DEVIATED SEPTUM & UVULECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
SURGERY* GUM SURGERY OUT PT (Surgical and medical procedures) | 0 (0) | 1 (2)
SURGERY* HERNIA (Surgical and medical procedures) | 1 (1) | 2 (2)
SURGERY* POSS BASAL CELL SKIN CANCER (Surgical and medical procedures) | 0 (0) | 1 (1)
SURGERY* PROSTATE RESTRUCTURING-ELECTIVE (Surgical and medical procedures) | 1 (1) | 0 (0)
SURGERY* RIGHT INGUINAL HERNIA REPAIR (Surgical and medical procedures) | 1 (1) | 0 (0)
SURGERY* ROTATOR CUFF REPAIR (Surgical and medical procedures) | 0 (0) | 1 (1)
SURGERY* TURP/HOSPITAL (Surgical and medical procedures) | 1 (1) | 0 (0)
SWELLING PERIPHERAL EDEMA (General disorders) | 1 (1) | 0 (0)
SWOLLEN ANKLES (PERIPHERAL EDEMA) (General disorders) | 1 (1) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
TINGLING BIL THIGH TO CALVES. OCCURS ~2X/MO (Nervous system disorders) | 0 (0) | 1 (1)
TINGLING IN FINGER TIPS (NEUROPATHYSENSORY) (Nervous system disorders) | 1 (1) | 0 (0)
TINNITUS (Ear and labyrinth disorders) | 12 (12) | 8 (11)
TINNITUS - SLIGHT INTERFERRENCE (Ear and labyrinth disorders) | 0 (0) | 1 (1)
TINNITUS CHRONIC (Ear and labyrinth disorders) | 0 (0) | 1 (1)
TINNITUS INCREASE (Ear and labyrinth disorders) | 0 (0) | 1 (1)
TINNITUS INCREASE, LEFT EAR (Ear and labyrinth disorders) | 0 (0) | 1 (1)
TINNITUS INCREASED (Ear and labyrinth disorders) | 0 (0) | 1 (1)
TINNITUS INCREASED, LEFT EAR (Ear and labyrinth disorders) | 1 (1) | 0 (0)
TINNITUS LEFT EAR (Ear and labyrinth disorders) | 0 (0) | 1 (1)
TINNITUS MAY HAVE INCREASED (Ear and labyrinth disorders) | 1 (1) | 0 (0)
TINNITUS MILD INCREASE, AUDIO AT 6M (Ear and labyrinth disorders) | 0 (0) | 1 (1)
TINNITUS PRE-EXISTING - INCREASED (Ear and labyrinth disorders) | 1 (1) | 0 (0)
TINNITUS VERY SLIGHT (Ear and labyrinth disorders) | 1 (1) | 0 (0)
TINNITUS X1 EPISODE (Ear and labyrinth disorders) | 1 (1) | 0 (0)
TINNITUS X4 EPISODES (Ear and labyrinth disorders) | 0 (0) | 1 (1)
TMJ (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
TOE INFECTION (Infections and infestations) | 0 (0) | 1 (2)
TOOTH ABCESS (Gastrointestinal disorders) | 1 (1) | 0 (0)
TOOTH INFECTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
TOOTH INFECTION -> ROOT CANAL (Gastrointestinal disorders) | 1 (1) | 0 (0)
UPPER HARD PALATE 1 CM ERYTHEMA W/ ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
UPPER RESPIRATORY INFECTION (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
URI (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (8)
URI CHEST CONGESTION/COUGH/PHLEGM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
URI COUGH AND SORE CHEST (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
URI SINUS INFECTION/COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
URI UPPER RESPIRATORY INFECTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
UTI (Renal and urinary disorders) | 9 (9) | 7 (8)
UTI (BACK PN) (Renal and urinary disorders) | 0 (0) | 1 (1)
UTI UTI SX (Renal and urinary disorders) | 0 (0) | 1 (1)
VERTIGO (Nervous system disorders) | 5 (5) | 1 (1)
VERTIGO POSITIONAL (Nervous system disorders) | 1 (1) | 0 (0)
VERTIGO SPINNING (Nervous system disorders) | 0 (0) | 1 (1)
VIRAL GASTROENTERITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
VISION (Eye disorders) | 0 (0) | 2 (2)
VISION BLURRED (Eye disorders) | 1 (1) | 0 (0)
VISION BLURRED RIGH EYE (Eye disorders) | 0 (0) | 1 (1)
VISION BLURRED WHEN READING (Eye disorders) | 0 (0) | 1 (1)
VISION BLURRING (Eye disorders) | 0 (0) | 1 (1)
VISION CATARACT (Eye disorders) | 1 (1) | 0 (0)
VISION CATARACT LEFT EYE (Eye disorders) | 0 (0) | 1 (1)
VISION CATARACTS, "FLASHING LIGHT" (Eye disorders) | 1 (1) | 0 (0)
VISION DISTURBANCE (Eye disorders) | 1 (1) | 0 (0)
VISION FLASHING LIGHTS - BILATERAL (Eye disorders) | 0 (0) | 1 (1)
VISION FLOATERS - LEFT EYE (Eye disorders) | 0 (0) | 1 (1)
VISION FLOATERS, RIGHT EYE (Eye disorders) | 1 (1) | 0 (0)
VISION GLAUCOMA (Eye disorders) | 1 (1) | 0 (0)
VISION INCREASED INTRAOCULAR PRESSURE (Eye disorders) | 0 (0) | 1 (1)
VISION LEFT EYE BLURRY (Eye disorders) | 0 (0) | 1 (1)
VISION MYOPIA, LACERATION (Eye disorders) | 0 (0) | 1 (1)
VISION RIGHT CATARACT (Eye disorders) | 0 (0) | 1 (1)
VISION SUB-CONJUNCTIVAL HEMMORHAGE (Eye disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 9 (9) | 5 (8)
VOMITING AND NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING NAUSEA AND VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITTING (Gastrointestinal disorders) | 0 (0) | 1 (1)
WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
WEAKNESS LEFT HAND (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
WEAKNESS LOWER EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
WEAKNESS NEW - LEFT ARM (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
WEAKNESS OVERALL (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
WEIGHT LOSS (Metabolism and nutrition disorders) | 10 (13) | 5 (5)
WEIGHT LOSS >5% (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
WEIGHT LOSS AND DIARRHEA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
WEIGHT LOSS DIETING (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
WEIGHT LOSS DURING RUN-IN PERIOD (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
WEIGHT LOSS INTENTIONAL (Metabolism and nutrition disorders) | 7 (7) | 4 (5)
WEIGHT LOSS ON DIET REGIMEN (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
WEIGHT LOSS PURPOSEFUL (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
WEIGHT LOSS R/T ATKINS DIET (10 LBS) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
WHEEZING W/ SWEATING SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
WOUND INFECT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WOUND* FACIAL CUT FROM FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
WOUND* HEAD LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
WOUND* HEAD LACERATION ON SCALP (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less